Evaluation of Investigational Daily Disposable Multifocal Contact Lenses Produced with Different Manufacturing Processes

Protocol CR-6418

Version: 2.0

Date: 10 February 2021

Investigational Products: JJVC Investigational Multifocal-PG Contact Lenses manufactured

in senofilcon A C3

Control: Dailies Total 1<sup>®</sup> Multifocal Contact Lenses manufactured in delefilcon A material

Keywords: Multifocal, Senofilcon A C3, Delefilcon A, Manufacturing, Presbyopia, Daily Wear, Daily Disposable, Dispensing, Randomized

## Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Council for Harmonization Good Clinical Practice E6(R2) (ICH GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

## **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| TABLE OF CO | ONTENTS |
|-------------|---------|
|-------------|---------|

| PROTO | OCOL TITLE, NUMBER, VERSION AND DATE | 6 |
|---|---|---|
| SPONS | OR NAME AND ADDRESS | 6 |
| MEDIC | CAL MONITOR | 6 |
| AUTHO | ORIZED SIGNATURES | 7 |
| CHANG | GE HISTORY | 9 |
| SYNOF | PSIS | 10 |
| | ONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF T | |
| | TRODUCTION AND BACKGROUND | |
| 1.1. | Name and Descriptions of Investigational Products | |
| 1.2. | Intended Use of Investigational Products | |
| 1.3. | Summary of Findings from Nonclinical Studies | |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 17 |
| 1.5.<br>Study | Relevant Literature References and Prior Clinical Data Relevant to Proposed of 18 | Clinica |
| 2. ST | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 18 |
| 2.1. | Objectives | 18 |
| 2.2. | Endpoints | 18 |
| 2.3. | Hypotheses | 19 |
| 3. TA | ARGETED STUDY POPULATION | 20 |
| 3.1. | General Characteristics | 20 |
| 3.2. | Inclusion Criteria | 20 |
| 3.3. | Exclusion Criteria. | 20 |
| 3.4. | Enrollment Strategy | 21 |
| 4. ST | UDY DESIGN AND RATIONALE | 22 |
| 4.1. | Description of Study Design | 22 |
| 4.2. | Study Design Rationale | 22 |
| 4.3. | Enrollment Target and Study Duration | 22 |
| 5. TE | EST ARTICLE ALLOCATION AND MASKING | 22 |
| 5.1. | Test Article Allocation | 22 |
| 5.2. | Masking | 23 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 23 |
| 6. ST | UDY INTERVENTION | 24 |
| 6.1 | Identity of Test Articles | 2/ |

| 6.2. | Ancillary Supplies/Products | 24 |
|-------|---------------------------------------------------|----|
| 6.3. | Administration of Test Articles | 25 |
| 6.4. | Packaging and Labeling | 25 |
| 6.5. | Storage Conditions | 25 |
| 6.6. | Collection and Storage of Samples | 25 |
| 6.7. | Accountability of Test Articles | 26 |
| 7. ST | UDY EVALUATIONS | 27 |
| 7.1. | Time and Event Schedule. | 27 |
| 7.2. | Detailed Study Procedures | 30 |
| VI | SIT 1 | 30 |
| VI | SIT 2 | 35 |
| VI | SIT 3 | 39 |
| VI | SIT 4 | 45 |
| VI | SIT 5 | 49 |
| VI | SIT 6 | 55 |
| FI | NAL EVALUATION | 57 |
| 7.3. | Unscheduled Visits | 58 |
| 7.4. | Laboratory Procedures | 59 |
| 8. SU | BJECTS COMPLETION/WITHDRAWAL | 59 |
| 8.1. | Completion Criteria | 59 |
| 8.2. | Withdrawal/Discontinuation from the Study | 60 |
| 9. PR | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 60 |
| 9.1. | Systemic Medications | 61 |
| 10. I | DEVIATIONS FROM THE PROTOCOL | 61 |
| 11. S | STUDY TERMINATION | 62 |
| 12. P | PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 63 |
| 13. A | ADVERSE EVENTS | 64 |
| 13.1. | Definitions and Classifications | 64 |
| 13.2. | Assessing Adverse Events | 66 |
| 13. | 2.1. Causality Assessment | 67 |
| 13. | 2.2. Severity Assessment | 67 |
| 13.3. | Documentation and Follow-Up of Adverse Events | 67 |
| 13.4. | Reporting Adverse Events | 69 |
| 13. | 4.1. Reporting Adverse Events to Sponsor | 69 |

| 13.4. | 2. Reporting Adverse Events to 70 | the Responsible IEC/IRB and Health Authorities |
|---|---|---|
| 13.5. | Event of Special Interest | 70 |
| 13.6. | Reporting of Pregnancy | 70 |
| . ST | ATISTICAL METHODS | 70 |
| 14.1. | General Considerations | 70 |
| 14.2. | Sample Size Justification | 71 |
| 14.3. | Analysis Populations | 71 |
| 14.4. | Level of Statistical Significance. | 72 |

Procedure for Handling Missing Data and Drop-Outs.......74

STUDY RECORD RETENTION.......81

PUBLICATION 82 REFERENCES 82

ETHICAL AND REGULATORY ASPECTS .......77

DATA HANDLING AND RECORD KEEPING/ARCHIVING......74

14.

14.5. 14.6.

14.7.

14.8.

14.9.

14.10.

15.1. 15.2.

15.3.

16.1.

16.2.

16.3.

16.4.

18.1.

18.2.

18.3.

18.4.

18.5.

19.

20.

21.

22.

15.

16.

17.

18.

| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIR | |
|---|---|
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | |
| APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | |
| APPENDIX F: OCULAR DOMINANCE | |
| APPENDIX G: LENS FITTING GUIDE | |
| APPENDIX H: CONTROL LENS FITTING GUIDE | |
| APPENDIX I: C-QUANT STRAYLIGHT MEASUREMENT | |
| APPENDIX J: VISIONIX CORNEAL TOPOGRAPHY AND WAVEFRONT | |
| APPENDIX K: | |
| , LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS | |
| , EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | |
| , DETERMINATION OF NEAR ADDITION | 183 |
| , NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE | |
| , LENS FITTING CHARACTERISTICS | 192 |
| , SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS | 198 |
| , DETERMINATION OF DISTANCE SPHEROCYLINDRIC REFRACTIVE ERROR | |
| , BIOMICROSCOPY SCALE | 206 |
| , DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION | |
| , DISTANCE LOGMAR VISUAL ACUITY MEASUREMINE PROCEDURE | |
| , PATIENT REPORTED OUTCOMES | 221 |
| , VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATESTING | |
| APPENDIX L: VWI-0081, GUIDELINES FOR COVID-19 RISK MITIGATION | 232 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 243 |
| LIST OF TABLES | |
| Table 1: Test Articles | 24 |
| Table 2: Ancillary Supplies | 25 |
| Table 3: Time and Events | 27 |
| Table 4: Disallowed systemic medications | 61 |
| Table 5: Examples of major and minor protocol deviations | 62 |
| Table 6: Binocular High Luminance High Contrast Visual Performance – 1-W Follow-up | |

#### LIST OF FIGURES

#### PROTOCOL TITLE, NUMBER, VERSION AND DATE

Title: Evaluation of Investigational Daily Disposable Multifocal Contact Lenses Produced with

Different Manufacturing Processes

Protocol Number: CR-6418

Version: 2.0

Date: 10 February 2021

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### **MEDICAL MONITOR**



The Medical Monitor must be notified by the clinical institution/site by e-mail or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

## **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, ISO 14155, ICH guidelines, and the Declaration of Helsinki.

| Author | See Electronic Signature Report | |
|---------------------|---------------------------------|------|
| | | DATE |
| Clinical Operations | | |
| Manager | See Electronic Signature Report | |
| | | DATE |
| Biostatistician | See Electronic Signature Report | |
| | | DATE |
| Data Management | See Electronic Signature Report | |
| | | DATE |

Medical Safety Officer

| Officer | See Electronic Signature Report | |
|----------|---------------------------------|---------|
| | | DATE |
| Reviewer | See Electronic Signature Report | D.A.TEL |
| | | DATE |
| | See Electronic Signature Report | |
| Reviewer | | DATE |

## **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section | Date |
|---|---|---|---|
| | | Number(s) Affected | |
| 1.0 | | Original Protocol | 21 Jan 2021 |
| 2.0 | | Section 7.1-removed corneal | 10 Feb 2021 |
| | | topography and wavefront procedure | |
| | | in time and events. | |
| | | Section 3.1-corrected typo referring to myopes in population description. | |
| | | Appendix A-added preference | |
| | | questionnaires at visit 5. | |

## **SYNOPSIS**

| Protocol Title | Evaluation of Investigational Daily Disposable Multifocal Contact Lenses Produced with Different Manufacturing Processes |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Phase 2 |
| Trial Registration | This study will be registered on ClinicalTrials.gov. |
| Test Article(s) | Investigational Product: JJVC Investigational Multifocal-PG |
| Test TittleTe(s) | Contact Lenses manufactured in senofilcon A C3 |
| | Control: Dailies Total 1 <sup>®</sup> Multifocal Contact Lenses |
| | manufactured in delefilcon A material |
| Wear and Replacement | Wear Schedule: The test lenses will be used on a daily |
| Schedules | disposable basis. |
| Schedules | ± |
| | Replacement Schedule: The lenses will be replaced after a day |
| 01: 4: | of wear. |
| Objectives | The objective of this study is to evaluate the visual |
| | performance (logMAR) and subjective vision responses of the |
| | JJVC Investigational Multifocal-PG Contact Lenses |
| | manufactured in senofilcon A C3 and compare the results to |
| | Dailies Total 1® Multifocal Contact Lenses manufactured in |
| | delefilcon A material. |
| Ctorder Endonsints | Duins and a sint 1 a MAD visual a suite accura |
| Study Endpoints | Primary endpoint: logMAR visual acuity scores |
| G: 1 D : | Secondary endpoint: CLUE vision scores |
| Study Design | This is a single-masked, 2×3 crossover, randomized- |
| | controlled, dispensing clinical trial. A total of approximately |
| | 70 hyperopic eligible subjects will be targeted to complete the |
| | study. The subjects will be randomized and fit (Visit 1) in a |
| | study lens and wear the lens for 3±1 day then undergo |
| | optimization (Visit 2) and wear the optimized pair for |
| | approximately 1 week (7±1 day). At the follow-up visit (Visit |
| | 3) the endpoints will be measured and subjects will be fit in |
| | the 2 <sup>nd</sup> study lens. The visits will be repeated wearing the 2 <sup>nd</sup> |
| | study lens (Visit 3 Fit/Visit 4 Optimization/Visit 5 Follow up). |
| | At Visit 5 the subjects will be fit in a new pair of lenses that |
| | match the same type and power they were dispensed at Visit 4, |
| | and wear the lenses for 1 week (7±1 day). At the follow-up |
| | visit (Visit 6) the endpoints will be measured and the subject |
| | will be exited from the study |
| | The primary endpoint will be logMAR visual acuity scores |
| | and the secondary endpoint will be CLUE vision scores. |
| | See the flow chart at the end of the synopsis table for the |
| | schematic of the study visits and procedures of main |
| | Schematic of the study visits and bloccutes of main |

| Sample Size | A total of approximately 80 eligible subjects will be enrolled |
|---|---|
| | with 70 subjects targeted to complete. |
| Study Duration | The study will last approximately 2 to 4 months. |
| Anticipated Study | Healthy male and female volunteers with presbyopia will be |
| Population | screened as per criteria outlined below. All volunteers will |
| | have baseline measurements taken to ensure eligibility. The |
| | baseline procedures will occur after informed consent has |
| | been obtained. Subjects will have medical and contact lens |
| | history recorded, baseline questionnaires completed, and |
| | refractive and anterior segment status determined. For a detail |
| | flowchart of procedures below. |

| Eligibility Criteria - |
|------------------------|
| Inclusion |

Potential subjects must satisfy all of the following criteria to be enrolled in the study

### Inclusion Criteria after Screening:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent.
- 4. Subjects must own a wearable pair of spectacles if required for their distance vision.
- 5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
- 6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

#### Inclusion Criteria after Baseline:

- 7. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D in each eye.
- 8. The subject's refractive cylinder must be  $\leq 0.75$  D in each eye.
- 9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 10. The subject must have distance best corrected visual acuity of  $20/20^{-3}$  or better in each eye.

| Eligibility | Criteria – |
|-------------|------------|
| Exclusion | |

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
- 5. A history of amblyopia, strabismus or binocular vision abnormality.
- 6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See Table 9.1 for further examples.
- 7. Use of any ocular medication, with the exception of rewetting drops.
- 8. History of herpetic keratitis.
- 9. History of irregular cornea.
- 10. History of pathological dry eye.
- 11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 13. Any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.

Exclusion Criteria after Baseline:

14. Clinically significant (Grade 3 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.

| | <ul><li>15. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.</li><li>16. Any current ocular infection or inflammation.</li><li>17. Any current ocular abnormality that may interfere with contact lens wear.</li></ul> |
|---|---|
| Disallowed | Use of any prescription or over-the-counter (OTC) |
| Medications/Interventions | medications that may affect contact lens wear. |
| | See section 9.1 for details regarding disallowed systemic medications. |
| Measurements and | logMAR Visual acuity and Subjective responses for vision |
| Procedures | using the CLUE questionnaire. |
| Microbiology or Other | None |
| Laboratory Testing | |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any serious adverse event (SAE) where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- | Non-Preserved Rewetting drops, lens cases, glass vials, saline, |
| Specific Materials | ETDRS light cabinet, 4 M logMAR charts, and Near logMAR charts. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |

Figure 1: Study Flowchart



# COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

Add Near addition; the additional power required for near vision correction

ADE Adverse Device Effect

ADHD Attention Deficit Hyperactivity Disorder AE Adverse Event/Adverse Experience

AO1DfA ACUVUE OASYS® 1-DAY with HydraLuxe<sup>TM</sup> TECHNOLOGY for

**ASTIGMATISM** 

AOfA ACUVUE OASYS® 2-WEEK for ASTIGMATISM

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience
COM Clinical Operations Manager
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

D Diopter

DMC Data Monitoring Committee
eCRF Electronic Case Report Form
EDC Electronic Data Capture
ESD Evelid Stabilized Design

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure

ICH The International Council for Harmonization

IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LASIK Laser-Assisted in Situ Keratomileusis

LogMAR Logarithm of Minimal Angle of Resolution

OD Right Eye
OS Left Eye
OU Both Eyes

PIG Patient Instruction Guide
PQC Product Quality Complaint
PRK Photorefractive Keratectomy
PRO Patient Reported Outcome

QA Quality Assurance

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

The purpose of this study is to evaluate the visual performance and subjective responses of the JJVC Investigational Multifocal Contact Lens using a different manufacturing lens hydration process. The lenses differ from previous prototypes by using a different lens hydration process form previous similar lens prototypes that have been evaluated. The lens hydration process used in this study for the test lenses is used in some marketed lenses that are manufactured by Johnson & Johnson Vision Care, Inc

### 1.1. Name and Descriptions of Investigational Products

Investigational Product: JJVC Investigational Multifocal-PG Contact Lenses manufactured in senofilcon A C3

Control: Dailies Total 1® Multifocal Contact Lenses manufactured in delefilcon A material.

## 1.2. Intended Use of Investigational Products

All lenses are intended to correct spherical refractive error and presbyopia. For this study both of the lenses will be worn as a daily disposable lens, with the lenses being discarded after a day of wear. The Lenses will be fit in a randomized fashion. After fitting, each subject will return for an optimization visit and then a follow-up. The sequence will then be repeated with the other study lens type and then the lens type worn at visit 5 will be re-worn for an additional 6-8 days. Each subject will wear each study lens type for approximately 16-24 days. In addition, approximately half of the subjects will wear the test lens, with the other half wearing control lens, for another 6-8 days for a total 22-32 days of lens wear.

#### 1.3. Summary of Findings from Nonclinical Studies

Not Applicable

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

Anticipated risks and adverse reactions with this lens are similar to those with other soft daily wear contact lenses used to correct presbyopia. A listing of examples of adverse reactions is found in the Section 13 of this protocol. The investigator should follow normal clinical guidelines regarding examination and care of subjects who participate in this trial. Refer to study lens package insert for additional details for the control lens and the Investigational Brochure (IB) for the Investigational lens. Both the study multifocal contact lenses are designed for the correction of refractive spherical refractive error and presbyopia. The investigational study contact lens is manufactured in senofilcon A C3 and the control lens is

manufactured in delefilcon A. Both of the lenses will be worn in a daily disposable wear modality. These lenses are not intended for extended wear in this study.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

| The Test lenses have been previously tested in clinical studies |
|---|
| was discontinued early by the Sponsor due to the COVID 19 pandemic. There were no Adverse Events reported in At the time of writing of this protocol studies and do not have a final clinical study report. A summary of the lens performance in studies and is provided below. |
| In 30 subjects completed the study per the protocol. The lenses displayed good clinical vision performance with binocular, high luminance, high contrast logMAR visual acuity of -0.057 and 0.091 at distance and near respectively. |
| There was one adverse event reported during the study. The subject experienced mild upper respiratory virus and did not receive any treatment for this event. The event resolved and the subject completed the study. The investigator considered the event to be not related to study article/procedure. |
| In41 subjects completed the study per the protocol. The lenses displayed good clinical vision performance with binocular, high luminance, high contrast logMAR visua acuity of -0.104 and 0.058 at distance and near respectively. |

There were no adverse events reported during the study.

For information about the control product refer to study lens package insert for additional details (APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) and the Investigational Brochure (IB) for the Investigational product.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

The objective of this study is to evaluate the visual performance (logMAR) and subjective vision responses of the JJVC Investigational Multifocal-PG Contact Lenses manufactured in senofilcon A C3 and compare the results to Dailies Total 1® Multifocal Contact Lenses manufactured in delefilcon A material.

#### 2.2. Endpoints

Primary Endpoint:

#### Visual Performance (logMAR)

Visual Performance will be assessed binocularly at each 1-week follow-up evaluation under high luminance high contrast conditions. At distance (4 meters), VA is assessed using ETDRS Charts; while near (40 cm) and intermediate (64 cm) assessments will be made using reduced

| Guillon-Poling charts. See | in Appendix I for details |
|---|---|
| regarding the collection of visual acuity (logMAR). | |

Secondary Endpoint:

#### Subjective Vision

Subjective vision will be assessed using the Contact Lens User Experience (CLUE<sup>TM</sup>) questionnaire at each 1-Week follow-up evaluation. CLUE<sup>TM</sup> is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE<sup>TM</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>TM</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.<sup>6</sup>

## Other Endpoints:

- CLUE<sup>TM</sup> Comfort
- CLUE<sup>TM</sup> Handling
- Lens Optimization Summary
- Mechanical Lens Fit
- Slit Lamp Findings

#### 2.3. Hypotheses

All primary and secondary hypotheses must be met in order to satisfy the objective of this study.

#### Primary Hypotheses

- 1. After approximately 1 week of wear in the optimized lenses, the distance, binocular, high luminance, high contrast visual performance of the Test lens will be non-inferior compared to that of the Control lens. A non-inferiority margin of 0.05 logMAR will be used.
- 2. After approximately 1 week of wear in the optimized lenses, the intermediate, binocular, high luminance, high contrast visual performance of the Test lens will be non-inferior compared to that of the Control lens. A non-inferiority margin of 0.05 logMAR will be used.
- 3. After approximately 1 week of wear in the optimized lenses, the near, binocular, high luminance, high contrast visual performance of the Test lens will be non-inferior compared to that of the Control lens. A non-inferiority margin of 0.05 logMAR will be used.

### Secondary Hypotheses

1. After approximately 1 week of wear in the optimized lenses, the overall quality of vision of the Test lens will be non-inferior compared to that of the Control lens. A non-inferiority margin of -5 CLUE points will be used.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Healthy male and female subjects who are habitual soft contact lens wearers will be recruited. Subjects will be at least 40 years of age and not older than 70 years of age. They will be hyperopic and have presbyopia.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all the following criteria to be enrolled in the study:

Inclusion Criteria after Screening:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent.
- 4. Subjects must own a wearable pair of spectacles if required for their distance vision.
- 5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
- 6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or, if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix E).

#### Inclusion Criteria after Baseline:

- 7. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D in each eye.
- 8. The subject's refractive cylinder must be  $\leq 0.75$  D in each eye.
- 9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 10. The subject must have distance best corrected visual acuity of 20/20<sup>-3</sup> or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

## Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
- 5. A history of amblyopia, strabismus or binocular vision abnormality.
- 6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See Table 9.1 for further examples.
- 7. Use of any ocular medication, with the exception of rewetting drops.
- 8. History of herpetic keratitis.
- 9. History of irregular cornea.
- 10. History of pathological dry eye.
- 11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 13. Any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.

#### Exclusion Criteria after Baseline:

- 14. Clinically significant (Grade 3 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 15. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.
- 16. Any current ocular infection or inflammation.
- 17. Any current ocular abnormality that may interfere with contact lens wear.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

### 4.1. Description of Study Design

This is a 6-visit, subject-masked, multi-site,  $2\times3$  crossover dispensing trial. Approximately 80 subjects will be enrolled with an aim of approximately 70 subjects to complete the study.

The study begins with an initial visit (Visit 1). If a subject is found to meet all eligibility criteria, they will be randomized to one of two lens wear sequences (Test/Control/Control or Control/Test/Test) in a bilateral fashion.

If the subject is dispensed study lenses at the initial visit, five additional visits will be conducted. The first follow-up visit (Visit 2) will occur 3±1 days after the initial visit. At Visit 2, subjects will undergo lens optimization if necessary. Subjects will wear the study lenses for 7±1 days and then will return for their second follow-up at Visit 3. At Visit 3, subjects will be dispensed their second study lens per the randomization schedule. Subjects will return for their first follow-up visit (Visit 4) 3±1 days after Visit 3, for lens optimization. Subjects will return for their second follow-up visit 7±1 days after Visit 4. At Visit 5, subjects will be dispensed their 3rd study lens per the randomization schedule and wear the lens for 7±1 days. The final visit will be the follow-up (Visit 6).

#### 4.2. Study Design Rationale

Crossover designs are a well-established study design in which subjects are exposed to multiple treatments during different time periods. A 2×3 bilateral crossover design was considered to be the optimal design since the study period is relatively short the design can be cost effective and more efficient comparisons between treatments can be made than compared to a parallel study since fewer subjects are required to achieve the same pre-specified statistical power. Each subject will act as their own control to reduce the influence of potential confounding factors such as age, gender and vision correction.

#### 4.3. Enrollment Target and Study Duration

Approximately 80 eligible subjects will be enrolled with the aim of approximately 70 to complete the study. The study will last approximately 2-4 months.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a 2×3 crossover design. A computer-generated randomization scheme will be used to randomly assign subjects, in blocks of 4, to one of the two possible lens wear sequences: Test/Control/Control or Control/Test/Test. The random scheme will be generated using the PROC PLAN procedure from Statistical Analysis System (SAS) Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment per the randomization list and not pre-select or assign subjects. The randomized assignment of

subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- O Subject meets all the inclusion / exclusion criteria
- o Subject history and baseline information has been collected.

## 5.2. Masking

This is a single-masked study with the subjects being masked. The term partial masking is being used as subjects will not be told any information regarding the optical designs of the lenses beyond that they are intended to correct for their refractive error and presbyopia, however there are slight differences in the tint of the lenses which is impossible to mask from the subject.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing.
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme if applicable

Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

## 6. STUDY INTERVENTION

## 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test | Control |
|---|---|---|
| Name | JJVC Investigational | Dailies Total 1® Multifocal |
| | Multifocal Contact Lens | Contact Lens |
| | Process A | |
| Manufacturer | Johnson & Johnson® Vision | Alcon |
| | Care, Inc. | |
| | | N/A |
| Lens Material | senofilcon A (C3) | delefilcon A |
| Nominal Base Curve | 8.35 mm | 8.5 mm |
| Nominal Diameter | 14.3 mm | 14.1 mm |
| Nominal Distance | +1.00 D to +4.00 D in 0.25 D | +1.00 D to +4.25 D in 0.25 D |
| Powers (D) | steps | steps |
| Nominal ADD Powers | LOW, MID, HI | LO, MED, HI |
| (D) | | |
| Water Content | 38% | 33% |
| Center Thickness | 0.07 mm | 0.09 mm@ -1.00 D |
| @ -3.00 D | @ -3.00 D | |
| Oxygen Permeability | 103 | 156 |
| (Dk) | | @ -3.00 D |
| Wear Schedule in | Daily Wear | Daily Wear |
| Current Study | • | |
| Replacement | Daily | Daily |
| Frequency | | |
| Packaging Form (vial, | Blister | Blister |
| blister, etc.) | | |

## 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Single-Use Preservative-Free Rewetting Solutions (any one of these three rewetting solutions options may be supplied) | | |
|---|---|---|---|
| Solution Name/Description | Eye-Cept <sup>®</sup> ScleralFil <sup>®</sup> LacriP | | |
| | | Saline Solution | |
| Manufacturer | Optics Laboratory | B&L | Menicon |
| Preservative | Non-Preserved | Non-preserved | Non-preserved |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the investigator and/or the sponsor.

### 6.4. Packaging and Labeling

The test articles will be packaged in blisters, as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:

#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

## 7. STUDY EVALUATIONS

## 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1<br>Screening,<br>Baseline, | Visit 2<br>Treatment 1<br>Follow-up 1 | Visit 3<br>Treatment 1<br>Follow-up 2 | Visit 4 Treatment | Visit 5<br>Treatment | Visit 6<br>Treatment |
|---|---|---|---|---|---|---|
| | Treatment | Optimization | Treatment 2 | Follow-up | Follow-up | Follow-up |
| | 1 | - | | 1 | 2 | 1 |
| | | | | Optimizati | Treatment 3 | |
| | | | | on | 3 | |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 3±1 | Day 7±1 | Day 7±1 |
| | | from V1 | from V2 | from V3 | from V4 | from V5 |
| | | | Day 0 | | | |
| Estimated Visit | 2.5 hours | 1.0 hour | 2.0 hour | 1.0 hour | 2.0 hour | 1.5 hour |
| Duration | | | | | | |
| Statement of | | | | | | |
| Informed | X | | | | | |
| Consent | W. | | | | | |
| Demographics Medical | X | | | | | |
| History/Concomit | X | | | | | |
| ant Medications | 74 | | | | | |
| Adverse Events | | | | | | |
| and Concomitant | | | | | | |
| Medications | | X | X | X | X | X |
| Review | | | | | | |
| Compliance | | X | X | X | X | X |
| Habitual Contact | X | | | | | |
| Lens Information | Λ | | | | | |
| Contact Lens | X | | | | | |
| History | A | | | | | |
| Wear Time and | | | | | | |
| Comfortable | X | | | | | |
| Wear Time with | | | | | | |
| Habitual lenses | | | | | | |
| Wear Time and Comfortable | | | | | | |
| Wear Time with | | X | X | X | X | X |
| Study lenses | | | | | | |
| Screening | | | | | | |
| Inclusion/Exclusi | X | | | | | |
| on Criteria | Α. | | | | | |
| on oncome | | | | | l | |

| 77: 11 C | 77' '4 1 | 771 0 | 777 3 | 77 4 | 77, 5 | 77' '4 ( |
|---|---|---|---|---|---|---|
| Visit Information | Visit 1 | Visit 2 Treatment 1 | Visit 3 Treatment 1 | Visit 4 Treatment | Visit 5<br>Treatment | Visit 6 Treatment |
| | Screening, Baseline, | Follow-up 1 | Follow-up 2 | 1 reatment 2 | reatment 2 | 3 |
| | Treatment | Optimization | Treatment 2 | Follow-up | Follow-up | Follow-up |
| | 1 | 1 | | 1 | 2 | 1 |
| | | | | Optimizati | Treatment | |
| | | | | on | 3 | |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 3±1 | Day 7±1 | Day 7±1 |
| Time Tom | Day 0 | from V1 | from V2 | from V3 | from V4 | from V5 |
| | | | Day 0 | | | |
| Estimated Visit Duration | 2.5 hours | 1.0 hour | 2.0 hour | 1.0 hour | 2.0 hour | 1.5 hour |
| Subject Reported | | | | | | |
| Ocular | X | X | X | X | X | X |
| Symptoms | | | | | | 12 |
| Baseline PRO | | | | | | |
| (CLUE and | | | | | | |
| MRD) | X | | | | | |
| Questionnaire | | | | | | |
| CLDEQ-8 | | | | | | |
| Questionnaire | X | | X | | X | X |
| Distance and | | | | | | |
| Near Entrance | X | X | X | X | X | X |
| Visual Acuity | 71 | 71 | | | 71 | 71 |
| Lens Removal | X | X | X | X | X | X |
| Subjective | A | A | | | 71 | 74 |
| Refraction and | | | | | | |
| Distance Visual | X | | | | | |
| Acuity | | | | | | |
| Near ADD | | | | | | |
| Determination | X | | | | | |
| Ocular | | | | | | |
| Dominance | X | | | | | |
| ADD Refinement | X | | | | | |
| Near Visual | | | | | | |
| Acuity | X | | | | | |
| Biomicroscopy | X | Х | X | X | X | X |
| Baseline | | | | | | |
| Inclusion/ | | | | | | |
| Exclusion | X | | | | | |
| Criteria | | | | | | |
| Continuance | | | X | | X | |
| | Х | x (if | X | x (if | X | |
| Lens Selection | Λ | modified) | | modified) | Λ | |
| Lens Insertion | X | X | X | X | X | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 |
|---|---|---|---|---|---|---|
| v isit illioilliation | Screening, | Treatment 1 | Treatment 1 | Treatment | Treatment | Treatment |
| | Baseline, | Follow-up 1 | Follow-up 2 | 2 | 2 | 3 |
| | Treatment | Optimization | Treatment 2 | Follow-up | Follow-up | Follow-up |
| | 1 | | | l<br>Optimizati | 2<br>Treatment | 1 |
| | | | | on | 3 | |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 3±1 | Day 7±1 | Day 7±1 |
| | | from V1 | from V2<br>Day 0 | from V3 | from V4 | from V5 |
| | | | Day 0 | | | |
| Estimated Visit | 2.5 hours | 1.0 hour | 2.0 hour | 1.0 hour | 2.0 hour | 1.5 hour |
| Duration | | | | | | |
| 10-Minute | | x (if | | x (if | | |
| Settling | X | modified) | | modified) | X | |
| Visual | | | | | | |
| Satisfaction / | | | | | | |
| Subjective | X | X | X | X | X | X |
| Acceptance | | | | | | |
| Study Lens | | | | | | |
| Distance and | | | | | | |
| Near Visual | X | X | X | X | X | X |
| Acuity | | | | | | |
| Distance Over | | | | | | |
| Refraction and | X | X | X | X | X | |
| Visual Acuity | | | | | | X |
| Subjective Lens | | | 37 | 37 | | |
| Fit Assessment | X | X | X | X | X | X |
| Lens Deposits | | | X | | X | X |
| Lens Wettability | | | X | | X | X |
| Binocular Over | | | X | | X | X |
| Refraction | | | A | | Λ | Λ |
| Compliance | | X | X | X | X | X |
| Follow-up PRO | | | | | | |
| (CLUE / MRD) | | X | X | X | X | X |
| Questionnaire | | | | | | |
| Visual | | | X | | X | X |
| Performance | | | | | | |
| Modifications | X | X | | X | | |
| Distance and | | | ** | ** | | |
| Near Exit Visual | X | X | X | X | X | |
| Acuity | | | | | | |
| Dispensing | X | X | X | X | X | |
| Criteria | *- | | v | v | ** | |
| Instructions | X | X | X | X | X | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 |
|---|---|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Treatment | Treatment | Treatment |
| | Baseline, | Follow-up 1 | Follow-up 2 | 2 | 2 | 3 |
| | Treatment | Optimization | Treatment 2 | Follow-up | Follow-up | Follow-up |
| | 1 | | | 1 | 2 | 1 |
| | | | | Optimizati | Treatment | |
| | | | | on | 3 | |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 3±1 | Day 7±1 | Day 7±1 |
| | | from V1 | from V2<br>Day 0 | from V3 | from V4 | from V5 |
| Estimated Visit | 2.5 hours | 1.0 hour | 2.0 hour | 1.0 hour | 2.0 hour | 1.5 hour |
| Duration | | | | | | |
| Schedule Follow- | | | v | v | | |
| up | X | X | X | X | X | |
| Final Evaluation | | | | | | X |

## 7.2. Detailed Study Procedures

#### VISIT 1

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline PRO (CLUE and MRD) performance. If the subject is not wearing their lenses they must be rescheduled.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. NOTE: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's age, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subject's medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
| 1.5 | Habitual Lens Duration of Wear/Days per week | Questions regarding the subject's duration of contact lens wear and the minimum number of days they wear their lenses per week. |

| 1.6 | Contact Lens History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). |
|---|---|---|
| 1.7 | Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses | Record the subject's wear time and comfortable wear time with their habitual contact lenses. |
| 1.8 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after |
| | | screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms are not required. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.9 | Baseline PRO<br>(CLUE and MRD)<br>and CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their habitual lenses using the PRO (CLUE and MRD) questions. |
| 1.10 | Ocular Symptoms | The subject will respond to a verbal openended symptoms questionnaire. |
| 1.11 | Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 1.12 | Lens Removal | Have the subject remove their habitual lenses and store in an approved storage solution. |
| 1.13 | Subjective<br>Refraction and<br>Distance Visual<br>Acuity | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. NOTE: Best distance visual acuity with sphero-cylindrical refraction must be at least 20/20 <sup>-3</sup> in each eye for the subject to be eligible in the study. |

| Near ADD Determination | The near reading addition will be determined using the binocular crossed cylinder | |
|---|---|---|
| | • | |
| Ocular Dominance | Determine the distance ocular dominance with the best distance correction in place using a +1.00-blur test. If the results are equivocal use the sighting dominance test to determine the dominant eye used for the study. | |
| ADD Refinement | Place the BCC result in the trial frame and refine the near prescription with trial lenses (or flippers) under binocular conditions. | |
| Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm. Record the near visual acuity OD, OS and OU at 40 cm. | |
| Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any of these slit lamp findings are Grade 3 or higher, the subject will be discontinued. If discontinued a final examination must be completed. | |
| | expedited, preservative-free rewetting drops may be instilled. | |
| Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If so, proceed to lens fitting. If subject is deemed to be ineligible after baseline, proceed to Final Evaluation and | |
| | Determination Ocular Dominance ADD Refinement Near Visual Acuity Biomicroscopy Eligibility after | Determination using the binocular crossed cylinder technique (BCC) at 40 cm. Determine the distance ocular dominance with the best distance correction in place using a +1.00-blur test. If the results are equivocal use the sighting dominance test to determine the dominant eye used for the study. ADD Refinement Place the BCC result in the trial frame and refine the near prescription with trial lenses (or flippers) under binocular conditions. Near Visual Acuity Using the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm. Record the near visual acuity OD, OS and OU at 40 cm. Biomicroscopy FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any of these slit lamp findings are Grade 3 or higher, the subject will be discontinued. If discontinued a final examination must be completed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. Eligibility after Baseline All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered eligible. If so, proceed to lens fitting. If subject is deemed to be ineligible after |

| Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|
| Step | Procedure | Details |
| 1.20 | Randomization | Record the randomization ID. |
| 1.21 | Lens Selection | Select the lens pair and power based on the randomization scheme, spherical equivalent refraction and fitting guide for each eye. Record the Test lens parameters (power and lot number). |

| | I | T |
|---|---|---|
| 1.22 | Lens Insertion | Subjects will insert the lenses themselves. If |
| | | the lens is uncomfortable, inspect for damage |
| | | and remove, reinsert or replace as necessary. |
| | | Damaged lenses will be stored in labeled vial |
| | | with sterile saline, and clearly differentiated |
| | | from the other worn lenses that will be |
| | | shipped back to the Sponsor. Complete the |
| 1 22 | I and Cattling | Product Quality Complaint form. |
| 1.23 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. |
| 1.24 | Determine Visual | |
| 1.24 | | Determine if the subject's vision is |
| | Satisfaction | acceptable with the lenses. Allow the subject |
| | | to look down a hallway or out of a window |
| | | for distance vision assessments, and for them |
| | | to read a book, magazine or similar for near |
| 1.25 | C. 1 I D' | vision. |
| 1.25 | Study Lens Distance | Measure the distance and near visual acuity |
| | and Near Visual | OD, OS and OU. Record the results. |
| | Acuity | N. J. J. STDDG 2000 G. C. J. J. |
| | | Note: Use the ETDRS 2000 Series Chart 1 or |
| | | 2 near card placed at 40 cm to measure the |
| 1.06 | D' . O | Near visual acuity |
| 1.26 | Distance Over- | Perform a distance over-refraction OD and |
| | Refraction and | OS using loose lenses outside of the |
| | Distance Visual | phoropter under ambient room illumination. |
| | Acuity | The distance over-refraction may also be |
| | | refined under binocular conditions. Record |
| | | the results. The results of the distance over- |
| | | refraction may also be checked for the impact |
| | | on near vision under monocular and/or |
| 1.07 | 3 K 1'C' | binocular conditions. |
| 1.27 | Modifications | If the subject reports unsatisfactory vision or |
| | | is unable to obtain 20/30 distance visual |
| | | acuity OU with the lenses, then a |
| | | modification must be attempted. If the |
| | | subject reports satisfactory vision with the lenses a modification is not required, however |
| | | at the Investigator's discretion and based |
| | | upon their findings on the measured visual |
| | | acuity and/or over- refraction the investigator |
| | | may make a modification. |
| | | Up to two attempts at modification are |
| | | permitted, if necessary, in order to achieve an |
| | | acceptable distance and near binocular |
| | | performance for the subject, and to enable |
| | | 1 - |
| | | them to wear that particular lens type. |

| 1.28 | Lens Fit Assessment | Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 1.22-1.27 will be repeated for each modification. Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). |
|---|---|---|
| 1.29 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. NOTE: The distance visual acuity must be at least 20/30 OU for the lenses to be |
| 1.30 | Dispensing Criteria | <ul> <li>dispensed.</li> <li>The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 1.31 | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> </ul> |

| | | Instruct the subject no cleaning or disinfecting solutions will be used for this |
|---|---|---|
| | | lens type. |
| | | If determined necessary by the |
| | | Investigator sterile non-preserved |
| | | rewetting drops may be dispensed to be |
| | | used as needed for dryness. |
| | | Subjects will be instructed to wear lenses |
| | | for a minimum of 6 hours a day, every |
| | | day during the study. |
| | | Subjects will be instructed to wear their |
| | | glasses when not wearing the study |
| | | lenses. |
| | | A patient instruction booklet will be |
| | | provided. |
| | | <u>NOTE</u> : In the event a lens is lost or damaged, the subject will return to the clinical site for |
| | | replacement. As much as reasonably |
| | | possible, a damaged lens and packaging should be returned to the clinical site (wet, if |
| | | possible) and then returned to the Sponsor. |
| | | If lens damage is present, complete the |
| | | Product Quality Complaint Form. The lens |
| | | will be stored in labeled vial with saline, and |
| | | clearly differentiated from the other worn |
| | | lenses that will be shipped back to the |
| | | Sponsor. |
| 1.32 | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 3±1 days. |
| | | NOTE TO A CHARLES |
| | | <u>NOTE</u> : To count the follow-up visit as a day |
| | | of wear the Subject must have worn the |
| | | study lenses for 6 hours prior to the visit. |

## VISIT 2

The subjects must present to Visit 2 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| Visit 2: Treatment 1 Follow-up 1 | | |
|----------------------------------|-----------|---------|
| Step | Procedure | Details |

| 2.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
|---|---|---|
| 2.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 2.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for |
| | | at least 6 hours per day. To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 2.4 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 2.5 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 2.6 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the |
| 2.7 | Distance Over-Refraction and Distance Visual Acuity | Near visual acuity Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results and distance visual acuity OD and OS. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |
| 2.8 | Determination of<br>Lens Optimization | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and |
| | | based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide and steps 1.22-1.27 in Visit 1 Fitting allowing for at least 10 minutes of settling time between each lens modification. |
|---|---|---|
| 2.9 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). |
| | | • The subject should not proceed to wear the lenses if any of the following is observed: |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> </ul> |
| | | • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). |
| | | <u>NOTE</u> : If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses, and complete the Final Evaluation forms. |
| 2.10 | Collection of unworn lenses (if | Collect unworn lenses returned by the subject when lens power has been optimized. |
| | applicable) | If lens power was not changed allow the subject to use the unworn lenses dispensed at Visit 1 and dispense enough lenses of the same power to last the subject until their next visit. |
| 2.11 | Lens Removal | The study lenses will be removed and discarded. |
| 2.12 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit<br>Lamp Classification Scales will be used to<br>grade the findings. |

| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
|---|---|---|
| 2.13 | Insertion of Study<br>Lenses | Dispense the subject a new pair of lenses that match the distance and ADD power of the lenses that were removed in Step 2.11 above. |
| 2.14 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. NOTE: The distance visual acuity must be at least 20/30 OU for the lenses to be |
| 2.15 | Dispensing Criteria | <ul> <li>dispensed.</li> <li>The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 2.16 | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> </ul> |

| | | <ul> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> </ul> |
|---|---|---|
| | | NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |
| 2.17 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 days. NOTE: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

## VISIT 3

The subjects must present to Visit 3 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 3: Treatment 1 Follow-up 2 | |
|---|---|---|
| Step | Procedure | Details |
| 3.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 3.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 3.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day. To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 3.4 | PRO (CLUE and MRD) and CLDEQ-8 Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO (CLUE and MRD) and lens preference questionnaires. |
| 3.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 3.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 3.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 3.8 | Visual Performance<br>Distance (4M)<br>Intermediate (64 cm)<br>Near (40 cm) | Binocular Visual performance will be recorded for the following: Distance, Bright Illuminance High and Low Contrast ETDRS Charts 4M-HC#3 and LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast |

| | | Near (40 cm) High Contrast and Low<br>Contrast |
|---|---|---|
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) High Contrast ETDRS Charts 4M-HC#6 Near, Dim Illuminance (with <u>Near</u> goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). |
| | | <ul> <li>Note:</li> <li>The room illuminance must be between 7.3 and 7.9 EV (394-597 lux).</li> <li>Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m²).</li> <li>Guillon-Poling, Near Chart Luminance Acceptable Range 10.8-11.1 EV (223-274 cd/m²).</li> <li>Do not use the Mesopic filter for Dim luminance (Dim luminance will</li> </ul> |
| 3.9 | Binocular Distance<br>Over-refraction and | Perform a binocular over-refraction and record the OD and OS results and distance |
| | Distance Visual Acuity | visual acuity. Note: No lens changes are allowed based on the over-refraction. |
| 3.10 | Lens Fit Assessment | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> </ul> |

| | | <u>NOTE</u> : If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses, and complete the Final Evaluation forms. |
|---|---|---|
| 3.11 | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject. |
| 3.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. NOTE: Lenses do not need to be stored in a refrigerator. |
| 3.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 3.14 | Continuance | Determine whether the subject is eligible to continue in the study based on the examination findings. |

| | Visit 3: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 3.19 | Lens Selection | Select the lens pair and power based on the randomization scheme, spherical equivalent refraction (measured at Visit 1 baseline) and fitting guide for each eye. Record the Test lens parameters (power and lot number). |
| 3.20 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the Product Quality Complaint form. |
| 3.21 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. |
| 3.22 | Determine Visual Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to |

| | | read a book, magazine or similar for near |
|---|---|---|
| 3.23 | Distance and Near<br>Entrance Visual<br>Acuity | vision. Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and |
| 3.24 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | OU. Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |
| 3.25 | Modifications | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted, if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 3.19-3.25 will be repeated for each modification. |
| 3.26 | Lens Fit Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. |
| 3.27 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be |

| | | recorded to the nearest letter OD, OS and OU. |
|---|---|---|
| | | <u>NOTE</u> : The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 3.28 | Dispensing Criteria | The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued. |
| | | Distance Snellen acuity equal to or<br>better than 20/30 OU |
| | | Subject must indicate that the vision is acceptable. |
| | | • Subject must indicate that the comfort of the lenses is acceptable. |
| | | Lenses must have an acceptable general lens fit. |
| 3.29 | Patient Instructions | <ul><li>Instruct the Subject the following:</li><li>The lenses will be worn on a daily wear basis.</li></ul> |
| | | Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed. |
| | | A new lens will be opened and worn each day. |
| | | Instruct the subject to bring back all unworn study lenses. |
| | | Instruct the subject no cleaning or disinfecting solutions will be used for this lens type. |
| | | If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. |
| | | Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study. |

| | | <ul> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> </ul> |
|---|---|---|
| | | NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |
| 3.30 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 3±1 days. NOTE: To count the follow-up visit as a day |
| | | of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

## VISIT 4

The subjects must present to Visit 4 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 4: Treatment 2 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 4.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 4.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses Wear Time | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 4.3 | Compliance | Record the subject's compliance with wearing the study lenses. |

| 4.4 | Ocular Samuetana | NOTE: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
|---|---|---|
| 4.4 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 4.5 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 4.6 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity |
| 4.7 | Distance Over-Refraction and Distance Visual Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results and distance visual acuity OD and OS. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |
| 4.8 | Determination of Lens Optimization | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted, if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide and steps 3.20-3.25 in Visit 3 Fitting allowing for at least 10 minutes of settling time between each lens modification. |

| 4.9 | Lens Fit Assessment | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>NOTE: If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses, and complete the Final Evaluation forms.</li> </ul> |
|---|---|---|
| 4.10 | Collection of<br>unworn lenses (if<br>applicable) | Collect unworn lenses returned by the subject when lens power has been optimized. If lens power was not changed allow the subject to use the unworn lenses dispensed at Visit 3 and dispense enough lenses of the same power to last the subject until their next visit. |
| 4.11 | Lens Removal | The study lenses will be removed and discarded. |
| 4.12 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 4.13 | Insertion of Study<br>Lenses | Dispense the subject a new pair of lenses that match the distance and ADD power of the lenses that were removed in Step 4.12 above. |
| 4.14 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |

| | | <u>NOTE:</u> The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
|---|---|---|
| 4.15 | Dispensing Criteria | The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued. |
| | | Distance Snellen acuity equal to or |
| | | better than 20/30 OU |
| | | Subject must indicate that the vision is |
| | | acceptable. |
| | | Subject must indicate that the comfort |
| | | of the lenses is acceptable. |
| | | Lenses must have an acceptable general |
| | | lens fit. |
| 4.16 | Patient Instructions | <ul><li>Instruct the Subject the following:</li><li>The lenses will be worn on a daily wear basis.</li></ul> |
| | | Only enough lenses will be dispensed to |
| | | the subject to wear for the required |
| | | number of days until their follow-up visit. |
| | | No additional lenses will be dispensed. |
| | | A new lens will be opened and worn each |
| | | day. |
| | | <ul> <li>Instruct the subject to bring back all<br/>unworn study lenses.</li> </ul> |
| | | Instruct the subject no cleaning or |
| | | disinfecting solutions will be used for this |
| | | lens type. |
| | | If determined necessary by the |
| | | Investigator sterile non-preserved |
| | | rewetting drops may be dispensed to be |
| | | used as needed for dryness. |
| | | • Subjects will be instructed to wear lenses |
| | | for a minimum of 6 hours a day, every |
| | | day during the study. |
| | | Subjects will be instructed to wear their |
| | | glasses when not wearing the study |
| | | lenses. |

| | | • Subjects will be instructed to bring their habitual contacts or spectacles to the next visit. NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |
|---|---|---|
| 4.17 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 days. |
| | | <u>NOTE</u> : To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

## VISIT 5

The subjects must present to Visit 5 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 5: Treatment 2 Follow-up 2 | |
|---|---|---|
| Step | Procedure | Details |
| 5.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 5.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 5.3 | Compliance | Record the subject's compliance with wearing the study lenses. |

| | | NOTE: Subjects must have worn lenses for |
|---|---|---|
| | | at least 6 hours per day |
| | | To be counted as a day of wear at this visit |
| | | the Subject must have worn the study lenses |
| | | for 6 hours prior to the visit. |
| 5.4 | PRO (CLUE and | The subject will evaluate the vision |
| | MRD) and CLDEQ- | characteristics, comfort characteristics, |
| | 8 Questionnaires | handling characteristics, and visual |
| | | symptoms of the study lenses using the PRO |
| | | (CLUE and MRD) lens preference |
| | | questionnaires. |
| 5.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended |
| | | symptoms questionnaire |
| 5.6 | Subjective | Record whether the subject's distance and |
| | Acceptance | near vision with the lenses is acceptable. |
| 5.7 | Distance and Near | Distance and near Snellen visual acuity will |
| | Entrance Visual | be measured for each eye with the study |
| | Acuity | contact lenses in place. |
| | | E |
| | | For near measures use the ETDRS 2000 |
| | | Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and |
| | | OU. |
| 5.8 | Visual Performance | Binocular Visual performance will be |
| | Distance (4M) | recorded for the following: |
| | Intermediate (64 cm) | Distance, Bright Illuminance |
| | Near (40 cm) | High and Low Contrast ETDRS Charts |
| | | 4M- HC#3 and LC#3 |
| | | Near, Bright Illuminance |
| | | Reduced Guillon-Poling Charts Intermediate |
| | | (64 cm) High Contrast and Low Contrast |
| | | Near (40 cm) High Contrast and Low |
| | | Contrast |
| | | Distance, Dim Illuminance (with <i>Distance</i> |
| | | goggles) |
| | | High Contrast ETDRS Charts 4M-HC#6 |
| | | _ |
| | | Near, Dim Illuminance (with <u>Near</u> goggles) |
| | | Reduced Guillon-Poling charts |
| | | High Contrast Intermediate (64 cm) and Near |
| | | (40 cm). |
| | | Note: |
| | | <ul> <li>The room illuminance must be</li> </ul> |
| | | between 7.3 and 7.9 EV (394-597 |

| 5.9 | Binocular Distance<br>Over-refraction and | <ul> <li>lux).</li> <li>Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m²).</li> <li>Guillon-Poling, Near Chart Luminance Acceptable Range 10.8- 11.1 EV (223-274 cd/m²).</li> <li>Do not use the Mesopic filter for Dim luminance (Dim luminance will be simulated by using the goggles)</li> <li>Perform a binocular over-refraction and record the OD and OS results and distance</li> </ul> |
|---|---|---|
| | Distance Visual Acuity | visual acuity. Note: No lens changes are allowed based on the over-refraction. |
| 5.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). |
| | | The subject should not proceed to wear the lenses if any of the following is observed: |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> </ul> |
| | | <u>NOTE</u> : If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses, and complete the Final Evaluation forms. |
| 5.11 | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject. |
| 5.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. NOTE: Lenses do not need to be stored in a refrigerator. |
| 5.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit<br>Lamp Classification Scales will be used to<br>grade the findings. |

| | | If the clearance of the fluorescein needs to be |
|------|-------------|-------------------------------------------------|
| | | expedited, preservative-free rewetting drops |
| | | may be instilled. |
| 5.14 | Continuance | Determine whether the subject is eligible to |
| | | continue in the study based on the |
| | | examination findings. |

| | Visit 5: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 5.19 | Lens Selection | Select the same lens pair and power that was dispensed at Visit 4. Record the Test lens parameters (power and lot number). |
| 5.20 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the |
| 5.21 | Lens Settling | Product Quality Complaint form. Allow the study lenses to settle for a minimum of 10 minutes. |
| 5.22 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. |
| 5.23 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 5.24 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |

| 5.25 | Lens Fit Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Iimbal exposure at primary gaze or with extreme eye movement; edge lift; excessive movement in primary and up gaze; or insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up. NOTE: If lens fit is unacceptable subject will be discontinued from the study. Remove |
|---|---|---|
| 5.26 | Distance and Near<br>Exit Visual Acuity | the lenses, and complete the Final Evaluation forms. Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. NOTE: The distance visual acuity must be at least 20/30 OU for the lenses to be |
| 5.27 | Dispensing Criteria | <ul> <li>dispensed.</li> <li>The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 5.28 | Patient Instructions | Instruct the Subject the following: |

- The lenses will be worn on a daily wear basis.
- Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit.
   No additional lenses will be dispensed.
- A new lens will be opened and worn each day.
- Instruct the subject to bring back all unworn study lenses.
- Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.
- If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.
- Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.
- Subjects will be instructed to wear their glasses when not wearing the study lenses.
- A patient instruction booklet will be provided.
- Subjects will be instructed to bring their habitual contacts or glasses to the next visit.

NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor.

| 5.29 | Schedule | The subject will be scheduled to return for |
|---|---|---|
| | Follow-up | their follow-up appointment in $7\pm 1$ days. |
| | | <u>NOTE</u> : To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

## VISIT 6

The subjects must present to Visit 6 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| Visit 6: Treatment 2 Follow-up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| 6.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 6.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 6.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 6.4 | PRO (CLUE and<br>MRD) and CLDEQ-<br>8 Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO (CLUE and MRD) questionnaires. |
| 6.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 6.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 6.7 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be |

| | | recorded to the nearest letter OD, OS and |
|---|---|---|
| 6.8 | Visual Performance<br>Distance (4M)<br>Intermediate (64 cm)<br>Near (40 cm) | OU. Binocular Visual performance will be recorded for the following: Distance, Bright Illuminance High and Low Contrast ETDRS Charts 4M- HC#3 and LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast Distance, Dim Illuminance (with Distance goggles) High Contrast ETDRS Charts 4M- HC#6 Near, Dim Illuminance (with Near goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). |
| | | <ul> <li>Note:</li> <li>The room illuminance must be between 7.3 and 7.9 EV (394-597 lux).</li> <li>Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m²).</li> <li>Guillon-Poling, Near Chart Luminance Acceptable Range 10.8-11.1 EV (223-274 cd/m²).</li> <li>Do not use the Mesopic filter for Dim luminance (Dim luminance will be simulated by using the goggles)</li> </ul> |
| 6.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. |
| 6.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: |

| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>NOTE: If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses, and complete the Final Evaluation forms.</li> </ul> |
|---|---|---|
| 6.11 | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject. |
| 6.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. NOTE: Lenses do not need to be stored in a refrigerator. |
| 6.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |

### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Exit Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best-corrected distance visual acuity (OD and OS) to the nearest letter. Note: This step is not necessary if the subject was exited due to screen failure. |

| Final Evaluation | | |
|---|---|---|
| Step | Procedure | Details |
| F.3 | Exit Slit Lamp Biomicroscopy (for subjects that are | FDA Slit Lamp Classification Scale will be used to grade the findings. |
| | discontinued early) | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. This step is not necessary if the subject was exited due to screen failure. |
| | | <b>Note</b> : This step is not necessary if the subject was exited due to screen failure, or if biomicroscopy was performed as part of the final follow-up visit procedures (i.e., immediately prior to the final evaluation). |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected, as appropriate:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Documentation of any test article dispensed or collected from the subject, if applicable.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| Unscheduled Visit | | |
|---|---|---|
| Step | Step Procedure Details | |
| U.1 | Reason for unscheduled visit | Indicate if the <u>only</u> reason for the visit is that the subject requires additional test articles. If the reason is other than resupply of previously dispensed lenses, specify the reason for the visit. |
| U.2 | Chief Complaints (if applicable) | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.3 | Adverse Events and<br>Concomitant<br>Medications Review<br>(if applicable) | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| U.4 | Entrance VA (if applicable) | Record the entrance distance visual acuity (OD, OS) to the nearest letter. |
| U.5 | Subjective Sphero-<br>cylindrical<br>Refraction (if<br>applicable) | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS). |
| U.6 | Slit Lamp<br>Biomicroscopy (if<br>applicable) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| U.7 | Dispensing (if applicable) | If the subject requires additional lenses to complete the wear period and is eligible to do so, provide additional lenses per the dispensing instructions given in the detailed study procedures. |
| U.8 | Exit Visual Acuity (if applicable) | Record the subject's exit distance visual acuity (OD, OS) to the nearest letter. |

**Note**: If the only reason for the unscheduled visit is that the subject requires additional test articles, only the dispensing information needs to be recorded.

## 7.4. Laboratory Procedures

Not Applicable

### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent.
- they are eligible.
- completed all study visits

### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject withdrawal of consent.
- Subject not compliant to protocol.
- Subject lost to follow-up.
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant).
- Subject develops significant or serious adverse events necessitating discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE).
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject missed any study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation

Additional subjects may be enrolled be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear.

### 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film. A summary of disallowed medications is shown in Table 4.

NOTE: Subjects who previously used these medications on a temporary basis must have ceased that medication at least 1 week prior to signing the informed consent.

Table 4: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Anticholinergics | Irritable bowel syndrome, Parkinson's disease, peptic ulcer, cystitis, nasal congestion, cold symptoms, overactive bladder, COPD | Bentyl, Spiriva, Atrovent, Hyosyne, Levsin, Symax Fastab, Symax SL, Homax SL, Cogentin, Transderm Scop, etc. |
| Oral Phenothiazines | Antipsychotic disorders (schizophrenia, mania) | Compazine, Mellarill,<br>Thorazine, Phenagran, etc. |
| Oral/Inhaled<br>Corticosteroids | Arthritis, colitis, asthma, bronchitis, allergic or inflammatory conditions | Cortisone, Prednisone,<br>Hydrocortisone, Medrol,<br>Kenalog, Flonase etc. |
| Oral Retinoids | Seborrhea, acne | Isotretinoin, Acitretin, Alitretinoin, etc. |
| Oral Tetracycline | Urinary Tract Infection, acne, chlamydia, gonorrhea | Sumcyin, Acitsite,<br>Achromycin V, etc. |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation". Deviations

that contradict the information contained in the Informed Consent/Assent forms will be considered Major Deviations.

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature.

Protocol waivers are prohibited.

Table 5 lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 5: Examples of major and minor protocol deviations

| Deviation category | Major deviation | Minor deviation |
|---|---|---|
| Out-of-window visit | Visit attended more than 2 days out of visit window defined in study procedures | Visit attended 2 or fewer days out of visit window defined in study procedures |
| Unanswered PRO questions | For questionnaires where data is related to a primary or secondary endpoint, more than 2 PRO questions are unanswered (i.e., left blank) in a single domain (i.e. vision). | For questionnaires where data is related to a primary or secondary endpoint, 2 or fewer PRO questions are unanswered (i.e., left blank). For questionnaires where data where data is not related to a primary or secondary endpoint, any PRO questions are unanswered (i.e., left blank). |

In the case of a major protocol deviation, the decision of whether or not the subject will be excluded from the Per-Protocol analysis population will be made at the time of cohort review.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.

- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device."

**Note**: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

**Note**: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) – An SAE is any adverse event that led to any of the following:

Death

- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Fetal distress, fetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device."

**Note 1**: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

**Note 2**: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.<sup>1</sup>

**Unanticipated Adverse Device Effect (UADE)** – A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related, unlikely related, possibly related, or related see definition in section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild, moderate, or severe see definition in section 0).
- Outcome not recovered or not resolved, recovering or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.
- Actions Taken none, temporarily discontinued, permanently discontinued, or other.

### 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

## 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system.

All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review form must be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate

health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

## 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

### 13.4.1. Reporting Adverse Events to Sponsor

### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

### 13.5. Event of Special Interest

None

#### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Summaries will be presented by study lens type (Test and Control) and will be performed separately by completion status (Safety Population, Per-Protocol Population or Intent-to-Treat Population).

### 14.2. Sample Size Justification

This study was designed and powered to demonstrate that the binocular high luminance high contrast, visual performance (logMAR) of the Test lens at distance (4 meters), intermediate (64 cm) and near (40 cm) after 1-week of lens wear is non-inferior to the Control lens. Historical data for the Test lens with respect to visual acuity is presented in the Table below.

Table 6: Binocular High Luminance High Contrast Visual Performance – 1-Week Follow-up

| Position | Lens | Mean | SD* | Minimum | Maximum |
|----------------------|---------|----------|---------|---------|---------|
| Distance (4 M) | Test | -0.07354 | 0.08265 | -0.2400 | 0.2400 |
| | Control | -0.05216 | 0.08397 | -0.2200 | 0.1600 |
| Intermediate (64 cm) | Test | -0.05455 | 0.08698 | -0.2600 | 0.2600 |
| | Control | -0.04216 | 0.08039 | -0.2400 | 0.2200 |
| Near (40 cm) | Test | 0.0667 | 0.10249 | -0.1000 | 0.4400 |
| | Control | 0.0790 | 0.00947 | -0.1600 | 0.3000 |

\*SD: Standard Deviation

### Visual Performance (logMAR)

Sample size calculation for Visual performance (logMAR) was carried out using Monte Carlo simulation methods using PROC IML. One-thousand boot strap samples were simulated based on the historical data in **Table 6** above for each Position separately. An interclass correlation of 0.8 between study periods was used. For this sample size calculation, we assumed that there was no period or sequence effect since the Test and Control have not be evaluated together in the same clinical study. For each replicated sample a linear mixed model was used; lens was included as the only fixed effect. A variance component (VC) covariance structure was used to model measurements from the same subject across study periods. Seventy subjects to complete provides >99% power to meet all primary hypotheses (Distance, Intermediate and Near) associated with visual performance.

The plan is to enroll 80 eligible subjects with a target completion of 70 subjects. During the enrollment period, the subject drop-out rate with be closely monitored, if an unexpectedly high dropout rate is observed, then the targeted total enrollment number maybe be increased accordingly to ensure that a minimum of 70 subjects complete the study.

#### 14.3. Analysis Populations

#### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

### **Intent-to-Treat (ITT) Population:**

All subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

## 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

#### 14.5. Primary Analysis

All primary analysis will be conducted on the Intent-to-Treat Population. A sensitivity analysis will be conducted on the Per-Protocol population.

### Visual Performance (logMAR)

Binocular, high luminance, high contrast visual performance (logMAR) will be analyzed using a linear mixed model. Sequence of lens wear, study period, lens type, distance (4 M, 64 cm and 40 cm), first order carryover effect and the lens by distance interaction will be included as fixed effects. Other characteristics including, age, gender and race and ADD power may be included when appropriate. Site will be included as a random effect (G-side). The covariance between residual errors from the same subject and distance across study periods will be modeled using either homogenous compound symmetry (CS) or unstructured (UN) covariance structure. The structure that returns the lowest finite-sample corrected Akaike's Information criterion<sup>7</sup> will be selected as the structure that best fits the model. The Kenward and Roger method<sup>8</sup> will be used for the denominator degrees of freedom.

Comparisons between the Test and Control lenses will be carried out at each distance (4 M, 64 cm and 40 cm) using 2-sided 95% confidence intervals constructed of least square means (LSM) differences (Test minus Control) at the 1-week follow-up evaluation.

#### Primary hypothesis 1:

The null and alternative hypothesis for binocular distance HLHC visual performance to test for non-inferiority of the Test lens relative to the Control lens is as follows:

$$H_o$$
:  $\mu_{Test} - \mu_{Control} \ge 0.05 \log MAR$   
 $H_A$ :  $\mu_{Test} - \mu_{Control} < 0.05 \log MAR$ 

Non-inferiority will be declared if the upper limit of the 95% confidence interval of the LSM difference between the Test and Control is below 0.05 logMAR. i.e.  $P(\mu_{Test} - \mu_{Control} < 0.05) \ge 0.975$ .
## Primary hypothesis 2:

The null and alternative hypothesis for binocular Intermediate HLHC visual performance to test for non-inferiority of the Test lens relative to the Control lens is as follows:

$$H_o$$
:  $\mu_{Test} - \mu_{Control} \ge 0.05 \log MAR$   
 $H_A$ :  $\mu_{Test} - \mu_{Control} < 0.05 \log MAR$ 

Non-inferiority will be declared if the upper limit of the 95% confidence interval of the LSM difference between the Test and Control is below 0.05 logMAR. i.e.  $P(\mu_{Test} - \mu_{Control} < 0.05) > 0.975$ .

## Primary hypothesis 3:

The null and alternative hypothesis for binocular near HLHC visual performance to test for non-inferiority of the Test lens relative to the Control lens is as follows:

$$H_o$$
:  $\mu_{Test} - \mu_{Control} \ge 0.05 \text{ logMAR}$   
 $H_A$ :  $\mu_{Test} - \mu_{Control} < 0.05 \text{ logMAR}$ 

Non-inferiority will be declared if the upper limit of the 95% confidence interval of the LSM difference between the Test and Control is below 0.05 logMAR. i.e.  $P(\mu_{Test} - \mu_{Control} < 0.05) \ge 0.975$ .

### 14.6. Secondary Analysis

#### **CLUE Vision**

CLUE vision scores at the 1-week follow-up will be analyzed using a linear mixed model adjusting for baseline values as a covariate. Sequence of lens wear, study period, lens type will be included as fixed effects. Other factors such as, race, gender or ADD power may be included in the model as covariates when appropriate. Site will be included as a random effect (G-side). The covariance between residual errors from the same subject across study periods will be modeled using either homogenous compound symmetry (CS) or unstructured (UN). The structure that returns the lowest finite-sample corrected Akaike's Information criterion<sup>7</sup> will be selected as the structure that best fits the model. The Kenward and Roger method, (Kenward and Roger, 1997)<sup>8</sup> will be used for the denominator degrees of freedom.

Comparisons between the Test and Control lenses at the 1-week follow-up evaluation will be carried out using two-sided 95% confidence intervals constructed for the least-square mean difference (Test minus Control).

## Secondary Hypothesis 1:

The null and alternative hypothesis for CLUE vision to test for non-inferiority of the Test lens relative the Control lens is as follows:

$$H_o$$
:  $\mu_{Test} - \mu_{Control} \le -5$   
 $H_A$ :  $\mu_{Test} - \mu_{Control} > -5$ 

Non-inferiority will be declared if the lower limit of the 95% confidence interval for the least-square mean difference is greater than -5. i.e.  $P(\mu_{Test} - \mu_{Control} > -5) \ge 0.975$ 

## 14.7. Other Exploratory Analysis

CLUE<sup>TM</sup> comfort and handling scores will be descriptively summarized for each timepoint and lens type.

Further exploratory analysis may be undertaken at the discretion of the study responsible clinician.

#### 14.8. Interim Analysis

An interim analysis will be conducted after at least 20 subjects have completed the study. The interim read will include descriptive summaries on all primary and secondary endpoints. Additionally, descriptive summaries on other objectives will also be provided including: CLUE<sup>TM</sup> Comfort, Handling, Lens Optimization Summary, Mechanical Lens Fit and Slit Lamp Findings. Listings on any adverse events, corneal infiltrates of other slit lamp findings may also be provided if necessary.

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 15 imputations.<sup>9</sup>

#### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

## 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using the BioClinica EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External data sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

# 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClincalTrials.gov.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

#### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

## 16.4. Data Monitoring Committee (DMC)

An independent Data Monitoring Committee (DMC) will be established to oversee the study. Members of DMC must be free of significant conflicts of interest (i.e., financial, intellectual, professional, or regulatory), and are experts in all scientific disciplines needed to interpret the data and ensure study participant safety.

During the conduct of the trial, responsibilities of the DMC will be to periodically review and monitor the incidence of adverse events, determine whether the basic study assumptions

remain valid, evaluate whether the overall integrity, scientific merit and conduct of the study remain acceptable, and make recommendations to the Sponsor. DMC meetings will be held quarterly until all subjects have completed the study. The DMC may also meet for an ad hoc review of data in the event that a UADE or other event is reported that may affect the outcome and/or continuation of the study.

The DMC will receive a data review package prior to the scheduled meeting. Data packages will include the following information/listings:

- Subjects enrollment and disposition information, such as
  - Number and Reason for Subject Early Withdrawal
  - o Number of subjects screened, randomized, early withdrawal, and complete
  - Number and Reason for Screen Failure
- Medical History
- Concomitant Medications
- Adverse Events
- Protocol Deviations
- Product Quality Complaints

Additional descriptive summary statistics of study endpoints may be provided per the DMC's requests. Unless otherwise specified, the masking of the treatment information will be maintained in the data prepared for the DMC.

Detailed information regarding the roles and responsibilities of the DMC for this study is provided in the Data Monitoring Committee Charter.

### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

#### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue

participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, section 4 of the ICH E6(R2) guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with section 8 of the ICH E6(R2) guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor

- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki, current ICH GCP<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

## 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>5</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- 6. Wirth RJ, et al. Development of the Contact Lens User Experience: CLUE Scales. *Optom Vis Sci.* 2016;93(8):801-808.
- 7. Keselman HJ, Algina J, Kowalchuk RK, Wolfinger RD. A Comparison of Two Approaches for Selecting Covariance Structures in the Analysis of Repeated Measures. *Communications in Statistics—Simulation and Computation*. 1998;27:591-604.
- 8. Kenward MG, Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997;53:983–997.
- 9. SAS Institute Inc: SAS® 9.4 Statements: Reference, Third Edition. Cary, NC: SAS Institute Inc; 2014.

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)



Protocol 6418



PRO SPECIFICATIO 2 Final 2021-02-09 



PRO SPECIFICATIO 2 Final 2021-02-09





Protocol 6418



PRO SPECIFICATIO 2 Final 2021-02-09





Protocol 6418

Confidential

















Confidential




**Protocol 6418** 






CR-6418, v 2.0

Protocol 6418



APPENDIX B: PATIENT INSTRUCTION GUIDE (TO BE PROVIDED SEPERATLEY)

APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

Dailies Total 1® Multifocal Contact Lenses

# Alcon

# DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lenses for Daily Disposable Wear

W900236420

Important: This package insert is effective as of December 2019 and applicable to the delefilcon A contact lenses described below. Please read carefully and keep this information for future use. This package insert is intended for the eye care professional, but should be made available to patients upon request. The eye care professional should provide the patient with appropriate instructions that pertain to the patient's prescribed lenses. Copies of this package insert are available without charge from Alcon by calling Customer Service at 1-800-241-5999 or download from our website at www.alcon.com. In addition, a Patient Instruction Booklet is available which is recommended to be given to patients.



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.

#### PRODUCT DESCRIPTION

DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lenses are made from a lens material that is 33% water and 67% (delefilcon A) polymer, a silicone containing hydrogel with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. Lenses contain the color additive copper phthalocyanine, a light blue tint, which makes them easier to see when handling.

#### **Lens Properties**

· Refractive Index hydrated:

· Light Transmittance: Oxygen Permeability (Dk):

93% (@ 610 nm, -1.00 D) 140 x 10<sup>-11</sup> (cm<sup>2</sup>/sec)(ml 0<sub>2</sub> /ml x mm Hg), measured at 35° C (intrinsic Dk-Coulometric

method)

33% by weight in normal saline · Water Content:

· Surface Water Content: > 80%

#### **Lens Parameters**

13 0 to 15 0 mm Diameter Range Spherical Power Range -20.00 to +20.00 D 8 0 to 9 2 mm Base Curve Bange

#### Lens Parameters Available<sup>1</sup>

#### DAILIES TOTAL1® (delefilcon A) spherical contact lenses

 Chord Diameter: Center Thickness:

14.1 mm 0.09 mm @ -3.00 D (varies with power)

· Base Curve: 8.5 mm

Powers

-0.50 to -6.00 D (0.25 D steps) -6.50 to -12.00 D (0.50 D steps) +0.50 to +6.00 D (0.25 D steps)

# DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses

· Chord Diameter:

14.1 mm · Center Thickness: 0.09 mm @ -3.00 D (varies with

· Base Curve:

+6.00 D to -10.00 D (0.25 D steps) Powers:

ADD: LO, MED, HI

NOTE: Hereafter, DAILIES TOTAL1® spherical contact lenses and DAILIES TOTAL1® Multifocal contact lenses will simply be referred to as delefilcon A contact lenses unless product distinction is necessary.

#### **ACTIONS**

When hydrated and placed on the cornea, delefilcon A contact lenses act as a refracting medium to focus light rays on the retina.

#### INDICATIONS (Uses)

DAILIES TOTAL1® (delefilcon A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

#### **CONTRAINDICATIONS (Reasons Not To Use)** DO NOT use delefilcon A contact lenses when any of the following exists:

- Inflammation or infection of the anterior chamber of the eve
- · Active disease, injury or abnormality affecting the cornea, conjunctiva, or evelids

- · Microbial infection of the eye
- · Insufficiency of lacrimal secretion (dry eye) that interferes with contact lens wear
- Corneal hypoesthesia (reduced corneal sensitivity)
- Use of any medication that is contraindicated or interferes with contact lens wear, including eye medications
- · Any systemic disease which may be exacerbated by or interferes with contact lens wear
- · Allergic reactions or ocular irritation of the ocular surfaces or adnexa that may be caused by or exaggerated by the wearing of contact lenses
- · Patient history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance or abnormal ocular response to contact lens wear
- · If eyes become red or irritated

#### WARNINGS

#### Advise patients of the following warnings pertaining to contact lens wear:

- · Problems with contact lenses and lens care products could result in serious injury to the eye. It is essential that patients follow their eye care professional's directions and all labeling instructions for proper use of lenses and lens care products. Serious eye problems, including corneal ulcers, can develop rapidly and lead to loss of vision.
- Daily wear lenses are not indicated for overnight wear, and patients should be instructed not to wear lenses while sleeping. Clinical study results have shown that the risk of serious adverse reactions is increased when contact lenses are worn overnight2.
- Studies<sup>2</sup> have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- · If a patient experiences eye discomfort, foreign body sensation, excessive tearing, vision changes, or redness of the eye, the patient should be instructed to immediately remove lenses and promptly contact his or her eye care professional. It is recommended that contact lens wearers see their eye care professional regularly as directed.

#### **PRECAUTIONS**

To prevent damage to the eyes or to the contact lenses, the following precautions should be taken:

#### Special Precautions for the Eye Care Professional

Due to the small number of patients enrolled in the clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently when selecting an appropriate lens design and parameters, the eye care professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, central and peripheral thickness and optic zone diameter.

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore the continuing ocular health of the patient and lens performance on the eye should be carefully evaluated on initial dispensing and monitored on an ongoing basis by the prescribing eye care professional.

- · Fluorescein, a yellow dye, should not be used while the lenses are on the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is recommended for in eye use prior to inserting lenses. Avoid dispensing saline from an aerosol can directly into the eye.
- Patients who wear contact lenses to correct presbyopia may not achieve the best possible corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Before leaving the eye care professional's office, the patient should be able to promptly remove their lenses or should have someone else available who can remove their lenses for them.
- Eve care professionals should instruct the patient to remove the lenses immediately if the eye becomes red or irritated.
- Routine eye examinations are necessary to help assure the continued health of the patient's eyes. Eye care professionals should make arrangements with the patient for appropriate follow-up visits. Alcon recommends that patients see their eve care professional once each year, or more often, as recommended by the eye care professional.

- · Diabetics may have reduced corneal sensitivity and thus are more prone to corneal injury and do not heal as quickly or completely as non-diabetics.
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly

#### Eye Care Professionals should carefully instruct patients about the following safety precautions:

#### **Handling Precautions**

- · Be sure that before leaving the eye care professional's office the patient is able to promptly remove lenses or have someone else available to remove them.
- Good hygiene habits help promote safe and comfortable lens wear. Always wash, rinse and thoroughly dry hands with a lint-free towel before handling lenses.
- . REMOVE A LENS IMMEDIATELY if an eye becomes red or irritated
- · Always handle lenses carefully. Never use tweezers or other sharp objects such as fingernails to remove lenses from the lens container unless specifically indicated for that use.
- Do not use if blister package is damaged or not sealed completely. This may result in product contamination which can lead to a serious eye infection.
- . Ensure that the correct lens for each eye is available. Shake the blister pack gently prior to opening. Remove the lens from the blister pack by carefully pouring the lens onto the palm of your clean hand. Ensure the lens is right side out. Inspect lenses prior to insertion. Do not insert damaged lenses.
- To insert lenses:
- Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses.
- Place a lens on the tip of your clean and dry right or left index finger, place the middle finger of the same hand close to lower eyelashes and pull down the lower eyelid.
- Use the fingers of the other hand to lift the upper eyelid. Place the lens directly on the eye (cornea) and gently roll
- finger away from the lens. Look down and slowly remove the hand, releasing the
- Look straight ahead and slowly remove the other hand, releasing the upper lid. Blink gently.
- To remove lenses:
  - Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses. Make sure hands are clean and completely dry.
  - Blink fully several times
  - While looking up, slide the lens down onto the white part of
  - Remove the lens by pinching gently between the thumb and forefinger. Do not pinch the eye tissue.
  - If the lens is difficult to grasp, dry fingers once more and try again. Do not use rewetting drops in this instance.
- If a lens decenters on the eye, it may be possible to recenter it by: Closing the eye and massaging the lens into place, or
  - Looking in the direction of the lens and blinking gently, or
  - Gently pushing the off-centered lens onto the cornea with light finger pressure on the edge of the upper or lower evelid.
- . If a lens tears in the eye it will feel uncomfortable. Advise wearers it is impossible to lose a contact lens or part of a contact lens behind the eye and to remain calm. Lens pieces may be removed by pinching them as for normal lens removal, carefully avoiding pinching the eye tissue. If the lens pieces do not seem to remove easily, rinsing with saline is recommended. If this does not help, the wearer should contact an eye care professional for assistance.

#### **Lens Wearing Precautions:**

- · Patients should never exceed the prescribed wearing schedule regardless of how comfortable the lenses feel. Doing so may increase the risk of adverse effects.
- The lens should move freely on the eye at all times. If the lens sticks (stops moving) on the eye, follow the recommended directions in the Care for a Sticking Lens section. If non-movement of the lens continues, the patient should be instructed to consult their eye care professional immediately.
- The eye care professional should be consulted about wearing lenses during water sports and water related activities. Exposure to water or other non-sterile liquids while wearing

contact lenses in activities such as swimming, water skiing, and hot tubs may increase the risk of ocular infection, including but not limited to *Acanthamoeba keratitis*.

- Never allow contact lenses to come into contact with non-sterile liquids (including tap water and saliva) as microbial contamination can occur, which may lead to permanent eye damage
- Eye irritation, infection, or lens damage may result if cosmetics, lotion, soap, cream, hair spray, deodorant, aerosol products or foreign particles come in contact with lenses.
- Environmental fumes, smoke, and vapors should be avoided in order to reduce the chance of lens contamination or physical trauma to the cornea.
- Lenses should be disposed of each day upon removal from the eve.
- Discard any lens which has become dehydrated or damaged.
   Replace with a sterile, fresh, new lens.
- Note the correct lens power for each eye to prevent getting them mixed up.
- Always carry spare lenses with you or have back-up spectacles available.
- Do not share lenses with anyone as this may spread micro-organisms which could result in serious eye health problems.
- Do not use lenses beyond their expiration date.

#### Other Topics to Discuss with Patients:

- Periodic eye examinations are extremely important for contact lens wearers. Schedule and conduct appropriate follow-up examinations to determine ocular response. Alcon recommends that patients see their eye care professional once each year or as recommended by the eye care professional.
- Certain medications may cause dryness of the eye, increased lens awareness, lens intolerance, and blurred vision or visual changes. These include, but are not limited to, antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness. Caution patients using such medications accordingly and prescribe proper remedial measures.
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.

# Who Should Know that the Patient is Wearing Contact Lenses:

- Patients should inform their health care practitioners that they are wearing contact lenses.
- Patients should inform their employers that they are wearing contact lenses. Some jobs may require the use of eye protection equipment or may require that contact lenses not be worm.

It is strongly recommended that patients be provided with a copy of the DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) Contact Lenses Patient Instruction Booklet available from Alcon and understand its contents prior to dispensing the lenses

#### **WATER ACTIVITIES**

# Do not expose contact lenses to water while wearing them. Warning:

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when showering or swimming, discard them and replace with a new pair. Ask the Eye Care Professional for recommendations about wearing lenses during any activity involving water.

#### ADVERSE EFFECTS

Patients should be instructed to check eyes regularly to make sure they look well, feel comfortable and vision is clear. Potentially serious complications are usually accompanied by one or more of the following signs or symptoms:

- Moderate to severe eye pain not relieved by removing the lens
- Foreign body sensation
- Excessive watering or other eye secretions including mucopurulent discharge
- · Redness of the eyes
- Photophobia (light sensitivity)
- Burning, stinging or itching or other pain associated with the eyes
- Comfort is less compared to when the lens was first placed on eve
- · Poor visual acuity (reduced sharpness of vision)
- Blurred vision, rainbows or halos around objects
- Feeling of dryness

#### WHAT TO DO IF A PROBLEM OCCURS

Patients should be instructed that if any of the above signs

or symptoms are noticed, he or she should:

- IMMEDIATELY REMOVE THE LENSES.
- If the discomfort or problem stops, discard the lens and replace it with a new one.
- If the discomfort or problem continues after removing lens(es) or upon insertion of a new lens, IMMEDIATELY remove the lens(es) and contact the eye care professional for identification of the problem and prompt treatment to avoid serious eye damage.
- The patient should be informed that a serious condition such as corneal ulcer, infection, corneal vascularization, or iritis may be present, and may progress rapidly. Less serious reactions such as abrasions, infiltrates, and bacterial conjunctivitis must be managed and treated carefully to avoid more serious complications.
- Additionally, contact lens wear may be associated with ocular changes that require consideration of discontinuation or restriction of wear. These include but are not limited to local or generalized corneal edema, epithelial microcysts, epithelial staining, infiltrates, neovascularization, endothelial polymegathism, tarsal papillary changes, conjunctival injection or iritis.

#### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of **DAILIES TOTAL1®** brand (delefilcon A) contact lenses, please notify: Alcon Medical Safety in the USA at 1-800-757-9780.

#### FITTING GUIDE AND PATIENT BOOKLET

Conventional methods of fitting contact lenses apply to delefilcon A contact lenses. For a detailed description of the fitting techniques, refer to the <code>DAILIES TOTAL1®</code> and <code>DAILIES TOTAL1®</code> **Multifocal** (delefilcon A) Contact Lenses *Professional Fitting and Information Guide*. Both the professional fitting guide and a patient instruction booklet are available free of charge from: Alcon Laboratories, Inc. 6201 South Freeway

Fort Worth, TX, USA 76134-2099

#### **LENS WEAR & REPLACEMENT SCHEDULES**

DAILY WEAR (less than 24 hours, while awake):

- To avoid tendency of the daily wear patient to over-wear the lenses initially, stress the importance of adhering to a proper, initial wearing schedule. Normal daily wear of lenses assumes a minimum of 6 hours of non lens wear per 24 hour period.
- It may be advisable for patients who have never worn contact lenses previously to be given a wearing schedule that gradually increases wearing time over a few days. This allows more gradual adaptation of the ocular tissues to contact lens
- The maximum daily wearing time should be determined by the eye care professional based upon the patient's physiological eye condition because individual responses to contact lenses vary. There may be a tendency for patients to over-wear the lenses initially. The eye care professional should stress the importance of adhering to the initial maximum wearing schedule. Studies have not been conducted to show that delefilcon A contact lenses are safe to wear during sleep, therefore patients should be advised to remove their lenses while sleeping. Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24 hour period. Optimum individual wearing schedule will vary.
- Delefilcon A contact lenses are intended to be worn once (daily disposable wear) and then discarded at the end of each wearing period. The patient should be instructed to start the next wearing period with a fresh new lens.

#### **EMERGENCY LENS CARE**

Cleaning and disinfection of daily disposable lenses is not recommended. The patient should be reminded to have replacement lenses or back-up spectacles available at all times.

#### CARE FOR A STICKING LENS

If the lens sticks (stops moving) or begins to dry on the eye, instruct the patient to apply several drops of a recommended lubricating solution (used in accordance with package labeling). The patient should wait until the lens begins to move freely on the eye before attempting to remove it. It is important that the patient wash and dry their hands thoroughly before removing the lens. If the lens continues to stick, the patient should IMMEDIATELY consult the eye care professional.

#### IN OFFICE USE OF TRIAL LENSES

Eye care professionals should educate contact lens technicians concerning proper use of trial lenses.

Each contact lens is shipped sterile in a blister pack containing phosphate buffered saline solution. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to ensure sterility, the blister pack

should not be opened until immediately prior to use. For fitting and diagnostic purposes lenses should be disposed of after a single use and not be re-used from patient to patient.

#### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should:

flush eyes immediately with tap water or fresh saline solution and immediately contact the eye care professional or visit a hospital emergency room without delay.

#### DISPOSAL AND RECYCLING

Dispose of contact lenses and the blister pack lidding in the waste bin, not down the sink or toilet. The carton packaging and the polypropylene (PP) plastic shell of the blister pack should be placed in the waste bin or recycled according to local waste management guidance.

#### HOW SUPPLIED

Each lens is packaged in a foil-sealed plastic container containing phosphate buffered saline solution with approximately 0.3% of polymeric wetting agents consisting of copolymers of polyamidoamine and poly(acrylamide-acrylic) acid and is steam sterilized. The package is marked with the base curve, diameter, dioptric power (and ADD power for multifocal lenses), manufacturing lot number, date of manufacture, and expiration date.

The following may appear on the labels or cartons:

#### Symbol/Abbreviation Description

| RX only | CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional. |
|---|---|
| | Single sterile barrier system |
| STERILE | Sterilized using steam |
| | Use-by date (Expiry date) |
| LOT | Batch code |
| en | Two letter code for the language (Example shown: English) |
| 2 | Do not re-use |
| 8 | Do not use if blister package is damaged |
| DIA | Diameter |
| BC | Base curve |
| PWR | Power |
| L | Left |
| R | Right |
| D | Diopter (lens power) |
| ADD | Addition power |
| MAX ADD | Maximum effective addition power |
| L0 | Low |
| MED | Medium |
| HI | High |
| C€ | European conformity mark |
| <u> </u> | Caution |
| (li | Consult instructions for use |
| EC REP | Authorized representative in the European Community |
| | Manufacturer |
| سا | Date of manufacture |
| MD | Medical device |
| 0 | Packaging waste license sign |

Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099

1-800-241-5999

www.alcon.com

U.S. Pat.: www.alconpatents.com

# Alcon

© 2019 Alcon Inc.

CR-6418, v 2.0

JJVC CONFIDENTIAL


<sup>&</sup>lt;sup>1</sup> Check for actual product availability as additional parameters may be introduced over time.

<sup>&</sup>lt;sup>2</sup>Schein, OD, Glynn RJ, Poggio EC, Seddon JM, Kenyon KR. The Relative Risk of Ulcerative Keratitis Among Users of Daily Wear and Extended Wear Soft Contact lenses. *N Eng J Med.* 1989; 321 (12):773-783.

# APPENDIX D: BINOCULAR OVER REFRACTION



APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE

| _ |
|---|
| _ |

APPENDIX F: OCULAR DOMINANCE



APPENDIX G: LENS FITTING GUIDE





APPENDIX H: CONTROL LENS FITTING GUIDE

# Professional Fitting and Information Guide

DAILIES TOTAL1\*
and
DAILIES TOTAL1\* Multifocal
(delefilcon A) Soft Contact Lenses
For Single-Use, Daily Disposable Wear

**Water Gradient One-Day Contact Lenses** 



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.



This page intentionally left blank

# **Table of Contents**

| Introduction | 5 |
|-----------------------------------------------------------|----|
| Product Description | 5 |
| Lens Properties | |
| Available Lens Parameters | 6 |
| Actions | 6 |
| Indications (Uses) | |
| Contraindications, Warnings, Precautions, Adverse Effects | 7 |
| Adverse Effect Reporting | |
| Fitting Guidelines (Spherical Lenses) | |
| Patient Selection | 8 |
| Pre-fitting Examination | |
| Trial Lens Evaluation | |
| Lens Base Curve Selection | |
| Initial Lens Power Selection | |
| Lens Fit Assessment | 9 |
| Final Lens Power Determination | |
| Fitting Guidelines (Multifocal Lenses) | |
| Pre-Fitting Examination | |
| Patient Selection | |
| Initial Lens Selection | |
| Initial Lens Fitting Evaluation | 14 |
| Initial Lens Visual Evaluation | |
| Fitting Procedures | |
| Fitting Guidelines (Monovision) | |
| Patient Selection | |
| Eye Selection | |
| Special Fitting Considerations | |
| Near Add Determination | |
| Trial Lens Fitting | |
| Adaptation | |
| Other Suggestions | 21 |
| Dispensing Visit | |
| Follow-Up Examinations | |
| Follow-up Examination Procedures | |
| Lens Handling Hints | |
| Lens Insertion | |
| Lens Removal | |
| Care for a Sticking Lens | |
| In Office Care of Trial Lenses | |
| Additional Information | |
| Vertex Distance Conversion Chart | |
| Product Package Insert | 20 |

This page intentionally left blank

#### Introduction

Thank you for prescribing DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) daily disposable soft contact lenses. The benefits of a high oxygen transmissible and wettable lens material with a state of the art manufacturing process are combined to make DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) lenses. This guide contains important information regarding fitting procedures and aftercare of the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) contact lens patient.

# Daily Disposability:

By eliminating the need for lens care, daily disposable lenses offer your patients a major advancement in wearing convenience. The next time you prescribe lenses consider the health and comfort benefits of beginning each wearing period with a new pair of fresh, sterile lenses that are worn once and then discarded.

# LightStream\* Lens Technology:

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses are made from a proprietary silicone hydrogel material with a water content of approximately 33% water. The use of process automation, precision glass and quartz molds and photolithographic edge forming help ensure every lens has the same crisp optics, smooth surface finish and consistent edge quality from lens to lens. Delefilcon A contact lenses are produced under strictly controlled process conditions and inspected to exacting quality tolerances. As a result, you can be confident your patients will experience consistent vision, comfort, and ease of handling every day.

## PRODUCT DESCRIPTION

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal soft contact lenses are made a silicone containing hydrogel that is approximately 33% water and 67% delefilcon A polymer with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. This structure enables a silicone hydrogel lens with a water gradient that has:

- Over 80% water at the surface of the lens to mimic the water content of the cornea.
- High level of oxygen transmissibility through the lens.
- Excellent overall comfort.

The lenses contain and release phosphatidylcholine (DMPC), a phospholipid found naturally in the tears. In addition, lenses contain the color additive copper phthalocyanine, a light blue tint which makes them easier to see when handling. The lenses are packaged in strips of 5 individual blisters containing buffered saline with approximately 0.3% of polymeric wetting agents consisting of copolymers of polyamidoamine and poly(acrylamide-acrylic acid).

# **Lens Properties**

Refractive Index (hydrated): 1.42

Light Transmittance: ≥ 93% (@610 nm, -1.00D)
 Oxygen Permeability (Dk): 140 x 10<sup>-11</sup> (cm²/sec)

(ml O<sub>2</sub>/ml x mm Hg), measured at 35°C,

(intrinsic Dk - Coulometric method)

Water Content 33% by weight in normal saline

• Surface Water Content ≥ 80%

#### Available Lens Parameters<sup>1</sup>

**DAILIES TOTAL1\*** (delefilcon A) Spherical contact lenses

Chord Diameter Available: 14.1 mm

• Center Thickness: 0.09 mm @ -3.00D (varies with power)

Base Curve: 8.5 mm

Powers Available: -0.50 to -6.00D (0.25D steps); -6.50 to

-12.00D (0.50D steps)

+0.50 to +6.00D (0.25D steps)

# DAILIES TOTAL1\* Multifocal (delefilcon A)

Chord Diameter: 14.1 mm

• Center Thickness: 0.09 mm @ -3.00D (varies with power)

Base Curve: 8.5 mm

Powers: -0.25 to -10.00D (0.25D steps); plano to

+6.00D (0.25D steps) ADD: LO, MED, HI

<sup>1</sup>Check for actual product availability as additional parameters may be introduced over time.

## **Actions**

When hydrated and placed on the cornea delefilcon A soft contact lenses act as a refracting medium to focus light rays on the retina.

#### INDICATIONS (USES)

**DAILIES TOTAL1\*** (delefilcon A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

**DAILIES TOTAL1\* Multifocal** (delefilcon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

See WARNINGS for information about the relationship between wearing schedule and corneal complications.

# CONTRAINDICATIONS, WARNINGS, PRECAUTIONS AND ADVERSE EFFECTS

For additional important prescribing and safety information, refer to the Package Insert that is printed in the back of this guide.

#### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of DAILIES TOTAL1\* or DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses, in the USA please **contact Alcon Medical Safety at** 1-800-757-9780.

## FITTING GUIDELINES

Please see the appropriate sections of this booklet that contain guidelines for spherical, multifocal and monovision fitting techniques.

# FITTING GUIDELINES (Spherical Lenses)

# 1. Patient Selection

The patient characteristics necessary to achieve success with DAILIES TOTAL1\* (delefilcon A) spherical lenses are similar to those for other spherical soft contact lenses. A thorough pre-fitting examination should be conducted to ensure the patient is a suitable candidate for soft contact lens wear.

The following procedures should be followed when fitting DAILIES TOTAL1\* (delefilcon A) spherical lenses. For additional tips on fitting the monovision patient refer to the section *Monovision Fitting Guidelines*.

# 2. Pre-fitting Examination

# A pre-fitting examination is necessary to:

- assess the patient's motivation, physical state and willingness to comply with instructions regarding hygiene and wear schedule
- make ocular measurements for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

# A pre-fitting examination should include:

- a thorough case history
- a spherocylindrical refraction
- keratometry
- · tear film assessment
- biomicroscopy

#### 3. Trial Lens Evaluation

#### A. Lens Base Curve Selection

A well-fitted lens provides good movement, centration and comfort. An optimal fit can be achieved for the vast majority of patients with the single 8.5 mm base curve.

#### B. Initial Lens Power Selection

The initial power selection should be as close as possible to the patient's prescription after taking into account spherical equivalent and vertex calculations, if necessary.

# Spherical Equivalent Calculation

To determine initial lens power, convert the spherocylindrical spectacle Rx to its spherical equivalent as follows:

Spherical Equivalent = Sphere power + 1/2 (Cylinder Power)
Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D

## **Vertex Distance Conversion**

If the spherical equivalent is greater than  $\pm$  4.00D, a vertex distance correction is necessary (see *Vertex Distance Conversion Chart*) to determine the lens power required at the corneal plane.

Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D

Vertex compensation: -4.75 (initial lens power)

#### C. Lens Fit Assessment

Allow the lenses to settle on the eyes for approximately 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate.

Evaluate the fit and movement of the lenses on the eye in primary and up gaze positions. The **Push-up Test**, as described below, is an additional test of the lens evaluation. The following guidelines will be helpful in fit evaluation:

#### Characteristics of a Well-fitted Lens

A well-fitted DAILIES TOTAL1\* (delefilcon A) spherical contact lens satisfies the following criteria:

- 1. Good centration and full corneal coverage in all fields of gaze.
- 2. **Sufficient lens movement to allow tear exchange** under the lens during a blink in primary or upward gaze.
- 3. Satisfactory Push-up Test
  - This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
  - A well fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- Good comfort and stable visual response (with over refraction).

# Characteristics of a Tight (Steep) Lens Fit

A tight or steep lens fit would display some or all of the following characteristics:

- Insufficient or no lens movement during a blink in primary or upward gaze.
- 2. Unsatisfactory Push-up Test
  - A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- Good centration.
- Good comfort.
- Fluctuating vision between blinks.

# Characteristics of a Loose (Flat) Lens Fit

A loose lens fit would display some or all of the following characteristics:

- 1. **Reduced comfort**, usually accompanied by lower lid sensation.
- Poor centration with limbal exposure on exaggerated eye movement.
- 3. Lens edge standoff.
- Excessive lens movement during the blink in primary or upward gaze.
- 5. Unsatisfactory Push-up Test
  - A loose fitting lens will move easily but may remain decentered or slip under the upper lid.
- 6. Vision may be blurred after the blink.

An inverted lens may mimic the characteristics of a loose lens. If any of

the above signs occur remove the lens and check to make sure it is not inverted.

# **General Fitting Tips**

- Trial fitting of the individual eye is recommended.
- A well fitting lens will show movement of 0.1 to 0.5 mm.

## D. Final Lens Power Determination

After the characteristics of a well fitted lens have been satisfied, conduct a **spherical over-refraction** to determine the proper lens power to be dispensed.

Example: Diagnostic lens: -4.50

Over-refraction: -0.25 Final lens power: -4.75

# FITTING GUIDELINES (Multifocal)

The **DAILIES TOTAL1\* Multifocal** (delefilcon A) soft contact lens is a progressive aspheric simultaneous vision soft contact lens, intended to correct presbyopia with or without additional ammetropia, available in three ADD powers; low (LO), medium (MED) and high (HI). For each lens the near and intermediate powers are concentrated primarily in the central portion of the optical zone while the distance power is contained in the surrounding portion. The continuous changes in power across the surface of the lens allow patients requiring a reading addition of up to + 3.00D to see clearly at far, intermediate, and near distances.

Achieving high success with DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses is dependent on several factors, including the patient's motivation, expectations and visual wearing environment, as well as your skill in optimizing the lens powers to balance binocular performance at distance and near. The information in this guide is designed to provide you with the tools to manage your presbyopic patients through each stage of the process from the initial case history to post-fitting follow-up.

# 1. Pre-fitting Examination

# A pre-fitting examination is necessary to:

- determine whether a patient is a suitable candidate for DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses
- make ocular measurements and assessments for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

# A pre-fitting examination should include:

- a thorough case history
- detailed assessment of patient's individual visual demands
- understanding of patient's objectives for lens wear and expectations
- a distance spherocylindrical refraction, near add determination and measurement of pupil diameter
- keratometry
- tear assessment
- biomicroscopy

Note: The importance of a thorough case history should not be underestimated. The information gained through careful listening and probing will help greatly in satisfying each patient's unique needs.

#### 2. Patient Selection

The eye care professional should weigh several factors when considering patient selection for a DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lens fitting. When fitting a lens intended to correct for presbyopia, it is especially important to evaluate the particular visual needs, objectives, lifestyle and expectations of the individual patient. Prospective candidates may include current contact lens wearers, former wearers, and persons with no previous wear history. For former wearers it is important to determine the cause for discontinuation.

There are two general categories of candidates based on anticipated usage: those who seek to wear their lenses as their principal means

of vision correction, and those who wish to integrate the use of their contact lenses with spectacles. The integrative user often seeks to wear their lenses for sports or other occasional activities while reverting to spectacles under poor lighting or otherwise demanding vision conditions. In general, even the part-time user does not require more than a few moments re-adaptation time following an interval of no lens wear.

While candidates with greater than 1.00 diopter of refractive error have often been thought of as better candidates than those with low error or emmetropia, this is a generalization that often does not hold true for a given individual. Success is influenced by many factors and the eye care professional is encouraged to offer DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses to all interested presbyopic patients who satisfy the standard requirements for soft contact lens wear.

To summarize patient selection, the characteristics of "ideal candidates" and those that will be more difficult to fit" are listed below:

#### Ideal Candidates

- Refractive cylinder < 1.00D.</li>
- Attainable visual demands that do not depend upon resolving very fine (smaller than 20/20 letters) details at *both* distance and near for extended periods while wearing DAILIES TOTAL1\* Multifocal contact lenses.
- Emphasis on tasks where it is advantageous to have objects simultaneously in focus over a large range of viewing distances.
- Expectations consistent with actual everyday visual demands.
- Motivated to wear lenses and understands that vision may not always be as sharp as with spectacles for some distances or lighting conditions.
- Unable to adapt to monovision correction.

## Less than Ideal Candidates

- Critical or very fine visual demands at both distance and near.
- Refractive cylinder 

  1.00D (any axis) in one or both eyes or against-the-rule refractive cylinder 

  1.00D in one or both eyes.
- Monocular distance acuities poorer than 20/20 with spherical equivalent refractive correction.
- Myopic anisometropia where the refractive error for one of the two eyes is low (≤1.50D) and has not been habitually corrected.
- Pupil size larger (> 4 mm) or smaller (<3 mm) than norm for presbyopic population under natural illumination conditions.
- Abnormal binocular sensory function (e.g., amblyopia or strabismus).
- Expectation to discard and never use spectacles again, including reading glasses, even for special tasks or viewing conditions.
- Highly satisfied monovision wearers.
- Any other contraindications to successful contact lens wear such as tear abnormality or lid margin disease.

#### 3. Initial Lens Selection

#### A. Initial Base Curve Selection

DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses are available in a single 8.5 mm base curve.

## **B. Initial Lens Power Selection**

Note: A careful maximum plus spherocylindrical refraction and nearpoint add determination should be conducted prior to selecting a DAILIES TOTAL1\* Multifocal (delefilcon A) trial lens. Autorefraction findings should be refined manually to rule out effects of instrument myopia and ensure proper control of residual accommodation.

The DAILIES TOTAL1\* Multifocal lens design makes selecting the initial lens power easy. You need only manipulate the distance power. The optimum starting point is with a power that is equal to or *more plus or less minus* than the vertex corrected spherical equivalent spectacle refraction.

#### C. Initial ADD Selection

Note: A careful nearpoint ADD determination should be conducted prior to selecting a DAILIES TOTAL1\* Multifocal (delefilcon A) trial lens

The DAILIES TOTAL1\* Multifocal (delefilcon A) 3 ADD SYSTEM allows personalized fitting for presbyopic patients. The table below makes initial ADD selection easy.

#### DAILIES TOTAL1\* MULTIFOCAL ADD SELECTION

| SPECTACLE ADD | BOTH EYES |
|----------------|-----------|
| Up to +1.25 | |
| +1.50 to +2.00 | MED |
| +2.25 to +2.50 | HI |

| Example 1: | OD | | os |
|-------------------------------------|------------------|--------|----------|
| Spherical Rx: | -4.50 -0.75 x 90 | | -4.00D |
| Spherical equivalent (least minus); | -4.75D | | -4.00D |
| Vertex corrected power: | -4.50D | | -4.00D |
| Spectacle Add: | | +0.75D | |
| Eye Dominance: | | OD | |
| Initial Trial Lens: | -4.50 LO | | -4.00 LO |

| Example 2: | OD | | os |
|---|---|---|---|
| Spherical Rx: | +4.25 -0.25 x 180 | | +4.00 D<br>-0.50 x 180 |
| Spherical equivalent (least minus): | +4.25D | | +3.75D |
| Vertex corrected power: | +4.50D | | +3.75D |
| Spectacle Add: | | +2.00D | |
| Eye Dominance: | | os | |
| Initial Trial Lens: | +4.50 MED | | +3.75 MED |

# 4. Initial Lens Fitting Evaluation

- a) Insert the lenses selected in Section 3 (above). If the exact power is not available, choose the next closest least minus/most plus lens power in your trial set.
- b) Allow the lenses to settle on the eyes for approximately 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate with the patient's tears.
- c) Evaluate the fit of the lenses on the eye. The **Push-up Test** as described below is an important part of the lens evaluation. The following guidelines will be helpful in evaluating the physical fit of the lens:

#### Characteristics of a Well-fitted Lens

A well-fitted DAILIES TOTAL1\* Multifocal (delefilcon A) contact lens satisfies the following criteria:

- Full corneal coverage and good centration (no limbal exposure).
   A lens that is decentered > 1 mm, particularly temporal, is less likely to give adequate vision.
- Lens movement of 0.1 to 0.5 mm should be present to allow tear exchange under the lens during a blink in primary gaze or upward gaze and to avoid variable vision.

# Push-up Test:

- This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
- A well fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- Good comfort.
- Acceptable visual acuity with over-refraction.

# Characteristics of a Tight (Steep) Lens Fit

A tight or steep fit should not be dispensed. If a lens fit is judged to be too steep a flatter lens (larger base curve), if available, should be evaluated. A tight or steep lens fit would display some or all of the following characteristics:

- Good centration.
- Insufficient or no lens movement during a blink in primary gaze or upward gaze.
- Excessive conjunctival drag (visible movement of the conjunctival vessels when the lens moves during a blink or during the push-up test). Note: presbyopes often have loose conjunctiva, some conjunctival movement is occasionally seen and may not be a sign of a tight fit. See Push-up Test below.
   Push-up Test:
  - A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- Good comfort.
- Blurred vision between blinks.

# Characteristics of a Loose (Flat) Lens Fit

If a lens fit is judged to be too flat a steeper lens (smaller base curve), if available, should be evaluated. A loose lens fit would display some or all of the following characteristics:

- Decentration.
- Excessive lens movement during the blink in primary or upward gaze.

#### Push-up Test:

- A loose fitting lens will move very easily, well beyond the limbus and possibly encroaching upon or going beyond the pupil. It will then return very quickly to its original position and often times return lower than its original position.
- Reduced comfort.
- Lens edge standoff.
- Blurred vision immediately after the blink.

# 5. Initial Lens Visual Evaluation

While lenses are settling, it is helpful to take the patient from the exam room to a "real-world" setting such as a room with an outside view. Once an acceptable fit has been achieved, the visual performance of the lenses may be evaluated. Visual acuity is tested at distance. If necessary, a spherical over-refraction should be performed using a trial frame or hand held lenses rather than a phoropter. This technique is essential when fitting multifocal lenses because it allows the patient to maintain the head posture and direction of gaze (relationship between eye and head) that he or she would naturally use during everyday tasks. This ensures that the visual performance of the lens is being assessed under conditions where the on-eye positioning matches that which will occur when the lens is being used, for example, for near work activities. In addition, pupil size will not be artificially increased

by the reduction in light associated with looking through the aperture of the phoropter cells, or decreased by proximal cues associated with the nearness of the instrument.

# 6. Fitting Procedures

<u>Step 1</u>. After the trial lenses have settled for approximately 10 minutes, measure distance acuity while the patient is viewing the chart binocularly (i.e., simultaneously with both eyes). Next, evaluate the patient's subjective impression of the near vision when trying to read typical everyday material (e.g., a newspaper, magazine, and cell phone). Lighting and reading distance should be what is normal for the patient.

<u>Step 2</u>. If distance or near vision is unsatisfactory, perform a **binocular distance** over-refraction, as follows. Use hand-held trial lenses and encourage plus. For example, if a Plano and +0.25D over-refraction yields the same results, use the +0.25D endpoint. Re-check visual acuity and visual quality as described in Step 1 above. If over-refraction is other than plano, go immediately to new trial lenses, keeping ADD the same.

<u>Step 3</u>. If distance and near vision are satisfactory, dispense lenses and remind patient to use good light when reading fine print or use additional reading glasses if needed. It is helpful to let the patient experience the lenses in their natural environment before further procedures for enhancing vision are performed.

<u>Step 4</u>. **Enhanced Near Vision.** If near vision is unsatisfactory, determine the dominant eye by the following method. Determine the eye with **greatest plus acceptance** by placing +1.50 handheld trial lens over each eye alternately while patient views in the distance with both eyes open. Consider the eye for which binocular vision blurs *least* with the +1.50 to be the non-dominant eye. Other methods to determine the dominant eye are appropriate.

<u>Step 4A:</u> Check the patient's binocular acuity with +0.50 over the non-dominant eye to determine if near vision is improved and distance vision is still acceptable. If so, place a new trial lens with the same ADD on the non-dominant eye, adjusting the distance power by +0.50.

| Enhanced near vision, Step A | | |
|---|---|---|
| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE (PLUS ACCEPTED) |
| Up to +1.25 | L | with additional +0.50 |
| +1.50 to +2.00 | MED | with additional +0.50 |
| +2.25 to +2.50 | HI | with additional +0.50 |

Next, re-check visual acuity and visual quality as described in Step 1 above. If satisfactory, dispense new distance lens power for the non-dominant eye. If near vision is still unsatisfactory, proceed to Step B:

Step 4B: If near vision is still unsatisfactory, adjust ADD as shown below.

| Enhanced near vision, Step B | | |
|---|---|---|
| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE (PLUS ACCEPTED) |
| Up to +1.25 | MED | MED |
| +1.50 to +2.00 | MED | • |
| +2.25 to +2.50 | • | MED |

Note: It is common to question the rather non-intuitive step we suggest for enhancing vision at near in the HI ADD range, where the suggestion is to "back off" to a MED ADD for the non-dominant eye, the same suggestion we make for enhancing distance vision (below). The reason for this is that after establishing (in Step A) that increasing plus is not helpful, the next most common reason for blur at near (or distance) is unacceptable ghosting that degrades the image quality. Backing down to the MED ADD in one eye can often relieve that and actually improve vision at near.

<u>Step 5</u>: Enhanced Distance Vision. If distance over-refraction did not improve visual acuity, adjust ADD according to the chart below.

| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT<br>EYE<br>(PLUS ACCEPTED) |
|----------------|--------------|----------------------------------------|
| +1.50 to +2.00 | LO | MED |
| +2.25 to +2.50 | H | MED |

# FITTING GUIDELINES (Monovision) Patient Selection

# A. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. Patients with reduced visual acuity, such as the amblyopic patient, may not be a good candidate for monovision.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it must be determined by trial whether this patient can function adequately with monovision. Monovision contact lens wear may not be optimal for such activities as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- driving automobiles (e.g., driving at night). Patients who cannot pass requirements for a driver's license with monovision correction should not drive with this correction. An additional over-correction can be prescribed to improve vision.

#### B. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with bifocal reading glasses. Each patient must understand that monovision, as well as other presbyopic contact lenses, or other alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision in straight-ahead and upward gaze that monovision contact lenses provide compared to spectacle bifocals.

# **Eye Selection**

Generally, the non-dominant eye is corrected for near vision. The following test for eye dominance can be used:

# A). Ocular Preference Determination Methods

- Method 1 Determine which eye is the "sight eye". Have the
  patient point to an object at the far end of the room. Cover
  one eye. If the patient is still pointing directly at the object,
  the eye being used is the dominant (sighting) eye.
- Method 2 Determine which eye will accept the added power for near with the least reduction in distance vision. Place a trial spectacle near ADD lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

#### B). Refractive Error Method

For anisometropic corrections, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

# C). Visual Demands Method

 Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

# Example:

A person who places copy to the left side of the desk will usually function best with the near lens on the left eye.

# Special Fitting Considerations

#### **Unilateral Lens Correction**

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens while a bilateral myope may require only a distance lens.

- Examples:
- Emmetrope: A presbyopic emmetropic patient who requires a +1.75 diopter ADD would have a +1.75 lens on the near eye and the other eye left without a lens.
- Bilateral myope: A presbyopic patient requiring a +1.50 diopter ADD who is -2.50 diopters myopic in the right eye and -1.50 diopters myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.
- Unilateral astigmat:
  - a) Emmetropic in one eye, astigmatic in the other

| Spectacle Rx | Potential Monovision Rx |
|---------------------|----------------------------|
| O.D. Plano | Uncorrected for distance |
| O.S1.00 -1.00 x 090 | +0.50 -1.00 x 090 for near |
| Add: +1.50 | |

b) Myopic in one eye, astigmatic in the other

| Spectacle RX | Potential Monovision RX |
|---------------------|--------------------------------|
| O.D1.50 | Uncorrected for near |
| O.S2.00 -1.75 x 090 | -2.00 -1.75 x 090 for distance |

#### **Amblyopia**

The amblyopic patient may not be a good candidate for monovision.

# **Astigmatism**

Patients with less than 1.50 diopters of astigmatism might be successfully fit in DAILIES TOTAL1\* (delefilcon A) spherical lenses.

- Determine which eye to use for the near prescription (see Eye Selection, A-C, above)
- Add the appropriate near add power to the spherical component of the astigmatic prescription for that eye.

Example: Spectacle Rx Potential Monovision Rx

O.D.: -2.50 -0.75 x 180 -2.50 -0.75 x 180 for distance

O.S.: -3.00 -1.75 x 165 -2.00 -1.75 x 165 for near

Add: +1.00

Dominant eye: O.D.

#### Near Add Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

# **Trial Lens Fitting**

A trial lens fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the directions in the *General Fitting Guidelines and Base Curve Selection* described earlier in the guide.

Case history and standard clinical evaluation procedures should be used to determine the suitability of monovision. Determine which eye is to be corrected for distance and which eye is to be corrected for near. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Immediately after the correct power lenses are in place, walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tasks are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to news print and finally smaller type sizes.

After evaluating the patient's performance under the above conditions, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a less favorable prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a few minutes or for several weeks. The longer these symptoms persist, the poorer the chance for successful adaptation. To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it is recommended that patients be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several

weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive under optimal driving conditions. After adaptation, and success with these activities, the patient should be able to drive under other conditions with caution.

# Other Suggestions

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Have supplemental spectacles to wear over the monovision contact lenses for specific visual tasks. This is particularly applicable for those patients who cannot meet driver's licensing requirements with a monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Success in fitting monovision can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of the clear near vision in straight ahead and upward gaze with monovision.

The decision to fit a patient with a monovision correction is most appropriately left to the eye care professional in conjunction with the patient after carefully considering the patient's needs. All patients should be supplied with a copy of the **Patient Instruction Booklet**, which contains important instructions for the monovision wearer. You can obtain copies of the instruction book by calling customer service **in the USA at (800) 241-5999.** 

#### **DISPENSING VISIT**

To help ensure patient success the following steps should be conducted with each patient, even if they have previously worn contact lenses. Even experienced wearers are prone to develop bad habits over time.

DAILIES TOTAL1\* brand (delefilcon A) lenses are supplied sterile in foil sealed blister pack containers. Open the foil pack by peeling back the foil lidding material and gently slide the lens out of the container with your finger, or pour the lens onto the palm of your clean hand.

Conduct the following steps with each patient, even if they have previously worn contact lenses:

# A. Verification of Lens Fit

Evaluate lens fit and visual response with the lens on the eye. The criteria of a well-fitted lens should be met and the patient's visual acuity should be acceptable. If not, the patient should be refitted with a more appropriate lens.

# B. Hygiene and Lens Handling Instructions

Good hygiene and proper lens handling are important factors in achieving safe, comfortable lens wear. Instruct the patient on hygiene and handling of lenses. Patients who are unable to place and remove lenses should not be provided with them.

# C. Lens Wear and Replacement Schedules (see Package Insert)

Prescribe and explain the daily disposable wear schedule. Explain that lenses are to be discarded after each daily wearing period. Determine the maximum suggested daily wearing period based on the patient's physiological eye condition. There may be a tendency for the patient to overwear their lenses initially. For some patients who have never worn contact lenses consider a wearing schedule that allows for a gradual increase in wearing time.

# D. Lens Care Directions (see Package Insert)

The lenses are not intended to be cleaned or disinfected and should be discarded after a single use. The eye care professional may recommend lens rewetting drops, as needed.

# E. Specific Instructions for Presbyopic Patients

Specific instructions, explanations and demonstrations are important for optimizing patient success with multifocal contact lenses. The following information and instructions have proven useful in advising patients who wear DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses.

- A contact lens that contains different powers for distance and near involves greater technological and optical complexity than does a bifocal or multifocal spectacle lens. This is because the contact lens moves with the eye, rather than having the eye move up and down while the lens remains suspended in a frame. While the contact lens therefore gives an unobstructed field of view and greater freedom regarding where to look, these advantages may mean that the sharpness of vision may not always be exactly the same as what would be experienced with spectacles.
- Although many individuals use DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses for full-time wear, it is not unusual to find that there may be some activities where one prefers to wear spectacles, or where the disadvantages associated with spectacles are outweighed by other issues. This is an entirely normal and natural response to the challenges presented by presbyopia.
- Situations where vision with multifocal contact lenses may be less sharp or otherwise "different" than what is experienced with spectacles often involve low illumination (e.g., a semi-dark room), reduced visibility (e.g., outdoor conditions of fog or heavy rain), or isolated sources of very bright light (e.g., headlights of an oncoming vehicle on a narrow country road). Patients should be instructed to make use of good light when reading fine print.
- Patients should be aware that it might be advisable to refrain from wearing their lenses while driving, flying an airplane or operating heavy machinery while wearing their lenses until they gain some experience with the lenses in a similar visual environment.
- Small changes in lens power can often make a significant difference in the quality of the vision experienced with multifocal contact lenses. Such changes can be best tailored to

individual needs and environmental conditions that the patient will personally encounter on a day-to-day basis. Confidence and assurance that such refinements, if needed, can be achieved are important for patient motivation during the initial period of lens wear.

#### F. Additional Instructions

# Review the Package Insert

Provide the patient with all relevant information and precautions on the proper use of the lenses that are prescribed.

Provide the Patient Instruction Booklet for DAILIES TOTAL1\*
 and DAILIES TOTAL1\* Multifocal (delefilcon A) Contact Lenses.
 Give the patient a copy of the Patient Instruction Booklet for DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses. Review the contents so the patient clearly understands the prescribed lens wear, care, and replacement schedule. In the USA you can obtain copies of the instruction book by calling Alcon customer service at (800) 241-5999.

# Follow-Up Examinations

Follow-up care is extremely important for continued successful contact lens wear. Follow-up care should include:

- Case history, including questions to identify any problems related to contact lens wear
- Management of specific problems, if any, and
- A review with the patient of the lens wearing schedule, replacement schedule and handling procedures.

#### Follow-up Examination Procedures

- Patients should be instructed to wear lenses prior to a follow-up examination.
- Record patient's symptoms, if any.
- Measure visual acuity monocularly and binocularly with the contact lenses in place.
- Perform an over-refraction to check for residual refractive error.
- With a biomicroscope, evaluate lens fitting.
- Remove the lenses and conduct a thorough biomicroscopic examination with fluorescein. Rinse eyes with saline before re-inserting lenses.
- Evert upper lids to determine condition of tarsal conjunctiva.
- Periodically perform keratometry and spectacle refractions. These results should be recorded to compare to the initial measurements.
- If any observations are abnormal, use professional judgment to manage the problem and restore the eye to optimal conditions. If visual requirements are not satisfied during any follow-up examination, the patient should be re-fitted with a more appropriate lens.

# LENS HANDLING HINTS Lens Insertion

• When about to place the lens on the eye, make sure the lens sits up on the placement finger. The finger should be dry so surface tension does

- not cause the lens to adhere to the finger.
- Check to see that the lens is right side out. A lens that is placed on the eye inside out may not feel comfortable or provide good vision.

One way to do this is to perform the 'taco test' by placing the lens between your thumb and index finger and squeeze the edges together gently.

- If the edges come together, the lens is right side out.
- If the edges turn outward, the lens is wrong side out. Carefully reverse it with your fingers.



Another way is to place the lens on the tip of your index finger and check its shape.

- If the edge appears bowl-shaped, it is right side out.
- If the edge has a lip or flares outward, it is wrong side out and must be reversed.
- Place the lens directly onto the cornea (placing it on the lower sclera can lead to the lens folding after a blink). While continuing to hold both lids in place, the patient should look down to seat the lens. The lids may then be released.



#### Lens Removal

- Wash hands thoroughly with soap that does not have any oils, lotions or perfumes.
- Carefully dry hands with a clean, lint-free towel.

It is important to remind patients to **dry their hands thoroughly** prior to removing their lenses. The surface of DAILIES TOTAL1\* brand lenses is designed to stay very wet and lubricious, or slippery while on the eye. If their fingertips are wet they are likely to slip across the surface of the lens making removal more difficult.

- Slide the lens off the cornea (down or to the side) onto the sclera. This
  produces a fold in the lens, which assists in removal. With the index finger
  and thumb, gently pinch the lens off the eye.
- Discard lenses.

# Care for a Sticking Lens

• In the unlikely event that the lens sticks (stops moving) or begins to dry on the eye, instruct the patient to apply several drops of a recommended lubricating solution (used in accordance with package labeling). The patient should wait until the lens begins to move freely on the eye before attempting to remove it. If the lens continues to stick, the patient should immediately consult the eye care professional.

#### IN OFFICE CARE OF TRIAL LENSES

Eye care professionals should understand and educate contact lens technicians concerning proper use of trial lenses.

- Each contact lens is shipped sterile in a sealed blister pack containing phosphate buffered saline with additives. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to insure sterility, the blister pack should not be opened until immediately prior to use.
- Delefilcon A lenses are for daily disposable wear only and should be discarded after a single use. The lenses should be disposed of after a single use and not be re-used from patient to patient.

# ADDITIONAL INFORMATION

For assistance with fitting or clinical questions regarding DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal contact lenses eye care professionals having questions or problems should contact Medical Information Systems in the USA at (800) 241-7468. To order DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal contact lenses contact your Alcon sales representative or call Customer Service, in the USA at (800) 241-5999.
## **VERTEX DISTANCE CONVERSION CHART**

For minus lenses, read left to right; for plus lenses, read right to left. (12 mm Vertex Distance)

| 1- | + | - | + | - | + | - | + |
|------|------|-------|-------|-------|-------|-------|-------|
| 4.00 | 3.87 | 7.50 | 6.87 | 12.00 | 10.37 | 19.00 | 15.50 |
| 4.25 | 4.00 | 7.62 | 7.00 | 12.50 | 10.75 | 19.25 | 15.62 |
| 4.50 | 4.25 | 7.75 | 7.12 | 12.75 | 11.00 | 19.25 | 15.75 |
| 4.75 | 4.50 | 7.87 | 7.25 | 13.00 | 11.25 | 19.75 | 16.00 |
| 5.00 | 4.75 | 8.00 | 7.37 | 13.50 | 11.50 | 20.00 | 16.12 |
| 5.12 | 4.87 | 8.12 | 7.50 | 13.75 | 11.75 | 20.25 | 16.25 |
| 5.37 | 5.00 | 8.25 | 7.62 | 14.00 | 12.00 | 20.50 | 16.50 |
| 5.50 | 5.12 | 8.50 | 7.75 | 14.25 | 12.25 | 20.75 | 16.62 |
| 5.62 | 5.25 | 8.75 | 8.00 | 14.75 | 12.50 | 21.00 | 16.75 |
| 5.75 | 5.37 | 9.00 | 8.25 | 15.00 | 12.75 | 21.25 | 17.00 |
| 5.87 | 5.50 | 9.25 | 8.37 | 15.50 | 12.75 | 21.75 | 17.25 |
| 6.00 | 5.62 | 9.50 | 8.62 | 15.75 | 13.25 | 22.25 | 17.50 |
| 6.12 | 5.75 | 9.75 | 8.75 | 16.25 | 13.50 | 22.50 | 17.75 |
| 6.37 | 5.87 | 10.00 | 9.00 | 16.75 | 13.75 | 23.00 | 18.00 |
| 6.50 | 6.00 | 10.25 | 9.12 | 17.00 | 14.00 | 23.50 | 18.25 |
| 6.62 | 6.12 | 10.50 | 9.25 | 17.25 | 14.25 | 23.75 | 18.50 |
| 6.75 | 6.25 | 10.75 | 9.37 | 17.62 | 14.37 | 24.25 | 18.75 |
| 6.87 | 6.37 | 11.00 | 9.62 | 18.00 | 14.50 | 24.75 | 19.00 |
| 7.00 | 6.50 | 11.25 | 9.75 | 18.12 | 14.75 | 25.00 | 19.25 |
| 7.12 | 6.62 | 11.50 | 10.00 | 18.50 | 15.00 | 25.50 | 19.50 |
| 7.37 | 6.75 | 11.75 | 10.25 | 18.75 | 15.25 | 26.00 | 19.75 |

This page intentionally left blank

#### Alcon a Novartis company

#### DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) Soft Contact Lenses for Daily Disposable Wear

900038292

PORTANT: This package insert is effective as of March 2016 and applicable to the detellicon A contact lenses described below. Please read carefully and keep this information for future use. This package insert is interesting, but should be made available to patients upon request. The eye care professional should provide the patient with appropriate instructions that pertain to the patient's prescribed insert. Deliver to provide the patient with appropriate instructions that pertain to the patient's prescribed insert. Deliver the patient patient is present patient. In addition, a Patientician Bookelist is available which is recommended to be given to patients. ded for the eye care insert are available without



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.

PRODUCT DESCRIPTION

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses are made from a lens material that is 33% water and 67% (delefilcon A) polymer, a silicone containing hydrogel with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. Lenses contain the color additive copper phthalocyanine, a light blue tint, which makes them easier to see when handling.

#### Lens Properties

- · Refractive Index hydrated: Light Transmittance: 93% (@ 610 nm, -1.00D)
- 140 x 10<sup>-11</sup> (cm<sup>2</sup>/sec)(ml 0<sub>2</sub> /ml x mm Hg), . Oxygen Permeability (Dk): measured at 35° C (intrinsic Dk-Coulometric
- method) . Water Content: 33% by weight in normal
- Surface Water Content: > 80%

#### Lens Parameters

Diameter Range 13.0 to 15.0 mm Soherical Power Range -20.00 to +20.00D Base Curve Range 8.0 to 9.2 mm

#### Lens Parameters Available

#### DAILIES TOTAL1\* (delefilcon A) spherical

- Chord Diamete
- 0.09 mm @ -3.00D (varies · Center Thickness: with power) . Base Curve: 8.5 mm
- -0.50 to -6.00D (0.25D · Powers: steps); -6.50 to -12.00D (0.50D steps) +0.50 to

+6.00D (0,25D steps)

#### DAILIES TOTAL1\* Multifocal (delefilcon A)

- Chord Diameter: 14.1 mm Center Thickness 0.09 mm @ -3.00D (varies
- with power) 8.5 mm +6,00D to -10,00D (0,25D

steps) ADD: LO, MED, HI NOTE: Hereafter, DAILIES TOTAL1\* spherical lenses and DAILIES TOTAL1\* Multifocal contact lenses will simply be referred to as delefilicon A contact lenses unless product distinction is necessary.

#### ACTIONS

When hydrated and placed on the cornea, delefilcon A contact lenses act as a refracting medium to focus light rays on the retina.

DAILIES TOTAL1\* (delefilcon A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-disease eyes with up to approximately 1,50 diopters (D) of astigmatism that does not interfere with visual acuity.

DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

## CONTRAINDICATIONS (REASONS NOT TO USE) DO NOT use delefilcon A contact lenses when any of the following exists: • Inflammation of

mation or infection of the anterior chamber of the eye

- · Active disease, injury or abnormality affecting the cornea, conjunctiva, or eyelic
- Microbial infection of the eve
- . Insufficiency of lacrimal secretion (dry eye) that interferes with contact lens wear

  Corneal hypoesthesia (reduced corneal sensitivity)
- Use of any medication that is contraindicated or interferes with contact lens wear, including eye medications
- Any systemic disease which may be exacerbated by or
- interferes with contact lens wear
  Allergic reactions or ocular irritation of the ocular surfaces or adnexa that may be caused by or exaggerated by the wearing of contact lenses
- Patient history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance or abnormal ocular response to contact lens wear
- eyes become red or irritated

#### WARNINGS

Advise patients of the following warnings pertaining to contact lens wear:

- . Problems with contact lenses and lens care products could result in serious injury to the eya. It is essential that patients follow their eye care professional's directions and all labeling instructions for proper use of lenses and lens care products. Serious eye problems, including corneal ulcers, can develop rapidly and lead to loss of vision.

  Daily wear lenses are not indicated for overnight wear, and
- patients should be instructed not to wear lenses while sleeping. Clinical study results have shown that the risk of serious adverse reactions is increased when contact lenses are worn overnight<sup>2</sup>.
  • Studies<sup>2</sup> have shown that contact lens wearers who are
- smokers have a higher incidence of adverse reactions than
- If a patient experiences eye discomfort, foreign body sensation, excessive tearing, vision changes, or redness of the eye, the patient should be instructed to immediately remove lenses and promptly contact his or her eye care professional. It is recommended that contact lens wearers see their eye care professional regularly as directed.

#### PRECAUTIONS

To prevent damage to the eyes or to the contact lenses, the following precautions should be taken:

regowing precautions should be taken: Special Precautions for the Eye Care Professional: Due to the small number of patients enrolled in the clinical investigation of lenses, all refractive powers, design configurations or lens parameters available in the lens material are not evaluated in significant numbers. Consequently when selecting an appropriate lens design and parameters, the eye care professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, central and peripheral thickness and optic zone diameter. The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore the continuing ocular health of the patient and lens performance on the eve should be carefully evaluated on initial dispensing and monit by the prescribing eye care professional. nitored on an ongoing basis

- Fluorescein, a yellow dye, should not be used while the lenses are on the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is recommended for in eye use prior to inserting lenses. Avoid
- dispensing saline from an aerosol can directly into the eye. Patients who wear contact lenses to correct presbyopia may not achieve the best possible corrected visual acuity for either far or near vision. Visual requirements vary with the Individual and should be considered when selecting the most appropriate ype of lens for each patient
- Before leaving the eye care professional's office, the patient should be able to promptly remove their lenses or should have
- someone dise available who can remove their lenses for them.
  Eye care professionals should instruct the patient to remove
  the lenses immediately if the eye becomes red or irritated.
- · Routine eye examinations are necessary to help assure the continued health of the patient's eyes. Eye care professionals should make arrangements with the patient for appropriate

follow-up visits. Alcon recommends that patients see their eye care professional once each year, or more often, as recommended by the eye care professional.

- Diabetics may have reduced corneal sensitivity and thus are more prone to corneal injury and do not heal as quickly or completely as non-diabetics, Visual changes or changes in lens tolerance may occur during
- pregnancy or use of oral contraceptives. Caution patients

## Eye Care Professionals should carefully instruct patients about the following safety precautions: Handling Precautions:

- Be sure that before leaving the eye care profes the patient is able to promptly remove lenses or have someone
- the patient is able to promptly remove lenses or have someone desa available to remove them. Good hygiene habits help promote safe and comfortable lens wear. Always wash, rinse and thoroughly dry hands with a limi-free tower before handling lenses. REMOVE A LENS IMMEDIATELY if an eye becomes red or
- Always handle lenses carefully. Never use tweezers or other sharp objects such as fingernalls to remove lenses from the lens container unless specifically indicated for that use.
- Do not use if blister package is damaged or not sealed completely. This may result in product contamination which can lead to a serious eve infection.
- Ensure that the correct lens for each eye is available. Shake tensure until the correct ents for each eye is available. Shake the bilster pack gently prior to opening. Remove the lens from the bilster pack by carefully pouring the lens onto the palm of your clean hand. Ensure the lens is right side out. Inspect lenses prior to insertion. Do not insert damaged lenses.
- - Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses.
  - Place a lens on the tip of your clean and dry right or left index finger, place the middle finger of the same hand close to lower eyelashes and pull down the lower eyeld. Use the fingers of the other hand to lift the upper eyelid.
  - Place the lens directly on the eye (cornea) and gently roll
  - finger away from the lens.

    Look down and slowly remove the hand, releasing the
  - ower lid.
  - Look straight ahead and slowly remove the other hand. releasing the upper lid.
    Blink gently.
- To remove lenses
  - Wash and rinse hands thoroughly and dry completely with a dean, lint free towel before handling lenses. Make sure hands are clean and completely dry.
     Blink fully several times.

  - While looking up, slide the lens down onto the white part
  - of the eye,
    Remove the lens by pinching gently between the thumb and forefinger. Do not pinch the eye tissue.
    If the lens is difficult to grasp, dry fingers once more and
- try again. Do not use rewetting drops in this instance.

   If a lens decenters on the eye, it may be possible to recenter it
  - Closing the eye and massaging the lens into place, or

  - Looking in the direction of the lens and blinking gently, or
     Gently pushing the off-centered lens onto the cornea with
    light finger pressure on the edge of the upper or lower eyelid,
- If a lens tears in the eye it will feel uncomfortable. Advise wearers it is impossible to lose a contact lens or part of a contact lens behind the eye and to remain calm. Lens pieces may be removed by pinching them as for normal lens removal, carefully avoiding pinching the eye tissue. If the lens pieces do not seem to remove easily, rinsing with saline is recommended if this does not help, the wearer should contact an eye care professional for assistance.

- Patients should never exceed the prescribed wearing schedule regardless of how comfortable the lenses feel. Doing so may crease the risk of adverse effects.
- increase the risk of adverse effects.

  The lens should move freely on the eye at all times, if the lens sticks (stops moving) on the eye, follow the recommended directions in the Care for a Sticking Lens section. If non-movement of the lens continues, the patient should be instructed to consult their eye care professional immediately.

- · The eye care professional should be consulted about wearing lenses during water sports and water related activities. Exposure to water or other non-sterile liquids while wearing contact lenses in activities such as swimming, water skiing, and hot tubs may increase the risk of ocular infection, including but not limited to Acanthamoeba keratitis.
- Never allow contact lenses to come into contact with non-sterile liquids (including tap water and saliva) as microbial contamination can occur, which may lead to permanent eye
- Eye irritation, infection, or lens damage may result if cosmetics, lotion, soap, cream, hair spray, deodorant, aerosol products or foreign particles come in contact with lenses.

  Environmental fumes, smoke, and vapors should be avoided in
- order to reduce the chance of lens contamination or physical trauma to the cornea.

  Lenses should be disposed of each day upon removal from the
- Discard any lens which has become dehydrated or damaged.
- Replace with a sterile, fresh, new lens.

  Note the correct lens power for each eye to prevent getting them mixed up.
- Always carry spare lenses with you or have back-up spectacles available.

  Do not share lenses with anyone as this may spread micro-organisms which could result in serious eye health problems
- Do not use lenses beyond their expiration date.

#### Other Topics to Discuss with Patients:

- Periodic eye examinations are extremely important for contact lens wearers. Schedule and conduct appropriate follow-up examinations to determine ocular response. Alcon recommends that patients see their eye care professional once
- each year or as recommended by the eye care professional.

  Certain medications may cause dryness of the eye, increased lens awareness, lens intolerance, and blurred vision or visual changes. These include, but are not limited to, antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness. Caution patients using such medications accordingly and prescribe proper remedial
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.

- Who Should Know that the Patient is Wearing Contact Lenses:

  Patients should inform their health care practitioners that they are wearing contact lenses.

  Patients should inform their employers that they are wearing
- contact lenses. Some jobs may require the use of eye protection equipment or may require that contact lenses not be

It is strongly recommended that natients be provided with a copy of It is storingly recommended that patients be provided with a copy the DallLies TOTAL1\* and DallLies TOTAL1\* Multifocal Contact Lenses (deeflicon A) Patient Instruction Booklet available from Alcon and understand its contents prior to dispensing the lenses.

#### ADVERSE EFFECTS

ADVERSE EFFECTS
Patients should be instructed to check eyes regularly to make sure they look well, feel comfortable and vision is clear. Potentially serious complications are usually accompanied by one or more of the following signs or symptoms:

• Moderate to severe eye pain not relieved by removing the lens
• Foreign body sensation
• Excessive watering or other eye secretions including

- mucopurulent discharge

  Redness of the eyes

  Photophobia (light sensitivity)
- . Burning, stinging or itching or other pain associated with the eyes

  Comfort is less compared to when the lens was first placed on
- Poor visual acuity (reduced sharpness of vision) Blurred vision, rainbows or halos around objects

#### WHAT TO DO IF A PROBLEM OCCURS

- WHAT TO DO IF A PROBLEM OCCURS
  Patients should be instructed that if any of the above signs or symptoms are noticed, he or she should:

   DMMEDIATELY REMOVE THE LENSES,

   If the discomfort or problem stops, discard the lens and replace it with a new one.

   If the discomfort or problem continues after removing lens(es) or upon insertion of a new lens, DMMEDIATELY remove the lens(es) and contact the eye care professional for identification of the newblem and remover treatment to
- for identification of the problem and prompt treatment to avoid serious eye damage.

  The patient should be informed that a serious condition such as corneal ulcer, infection, corneal vascularization, or

iritis may be present, and may progress rapidly. Less serious reactions such as abrasions, infiltrates, and bacterial conjunctivitis must be managed and treated carefully to avoid more serious complications.

Additionally, contact lens wear may be associated with ocular

changes that require consideration of discontinuation or restriction of wear. These include but are not limited to local or restriction of wear. These induced but are not immed to local or generalized corneal edema, epithelial microcysts, pothelial staining, infiltrates, neovascularization, endothelial polymegathism, tarsal papillary changes, conjunctival injection

#### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of **DAILLES TOTAL1\*** brand (delefilcon A) contact lenses, please notify: Alcon Medical Safety in the USA at 1-800-757-9780.

#### FITTING GUIDE AND PATIENT BOOKLET

Conventional methods of fitting contact lenses apply to deleflicon A contact lenses. For a detailed description of the fitting techniques, refer to the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal Contact Lenses (delefficon A) Professional Fitting and Information Guide, Both the professional fitting guide and a patient instruction booklet are available free of charge from:

Alcon Laboratories, Inc.

6201 South Freeway Fort Worth, TX, USA 76134-2099 1-800-241-5999

#### LENS WEAR & REPLACEMENT SCHEDULES

- DAILY WEAR (less than 24 hours, while awake):
  To avoid tendency of the daily wear patient to overwear the lenses initially, stress the importance of adhering to a proper, initial wearing schedule. Normal daily wear of lenses assumes
- a minimum of 6 hours of non lens wear per 24 hour period, It may be advisable for patients who have never worn contact lenses previously to be given a wearing schedule that gradually increases wearing time over a few days. This allows more gradual adaptation of the ocular tissues to contact lens wear.
  - The maximum daily wearing time should be determined by the eye care professional based upon the patient's physiological eye condition because the patients physiological by contact lenses vary. There may be a tendency for patients to overwear the lenses initially. The eye care professional should stress the importance of adhering to the initial maximum wearing schedule. Studies have not been conducted to show that deleficon A contact lenses are safe to wear durin sleep, therefore patients should be advised to remove their lenses while sleeping. Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24 hour period. Optimum individual wearing schedule will vary.
- Delefilcon A contact lenses are intended to be worn once (daily disposable wear) and then discarded at the end of each wearing period. The patient should be instructed to start the next wearing period with a fresh new lens.

#### **EMERGENCY LENS CARE**

Cleaning and disinfection of daily disposable lenses is not recommended. The patient should be reminded to have replacement lenses or back-up spectacles available at all times.

#### CARE FOR A STICKING LENS

CARE FOR A STICKING LENS
If the lens sticks (stops moving) or begins to dry on the eye, instruct
the patient to apply several drops of a recommended lubricating
solution (used in accordance with package labeling). The patient
should wait until the lens begins to move freely on the eye before
attempting to remove it. It is important that the patient wash and
dry their hands thoroughly before removing the lens. If the lens
continues to stick, the patient should IMMEDIATELY consult the eye
ever professions.

## IN OFFICE USE OF TRIAL LENSES

Eve care professionals should educate contact lens technicians

Eye date protessiones amount outcome commentation concerning proper use of trial lenses.

Each contact lens is shipped sterile in a bilster pack containing phosphate buffered saline solution. Hands should be thoroughly washed and rinsed and dried with a fint-free towel prior to handling a lens. In order to ensure sterility, the bilster pack should not be opened until immediately prior to use. For fitting and diagnostic purposes lenses should be disposed of after a single use and not be re-used from patient to patient.

#### EMERGENCIES

The patient should be informed that if chemicals of any kind

Interplaced should be informed until inclinations or any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: Flush eyes immediately with tap water or fresh saline solution and immediately cortact the eye care professional or visit a hospital emergency room without delay.

#### HOW SUPPLIED

Each lens is packaged in a foil-sealed plastic container containing phosphate buffered saline solution with approximately 0.3% of polymeric wetting agents consisting of copolymers of polymeric wetting agents consisting of copolymers of polymidoamine and poly(acrylamide-acrylic) acid and is steam sterlized street . The package is marked with the base curve. diameter, dioptric power and ADD power (multifocal lenses) manufacturing lot number and expiration date

The following may appear on the labels or cartons:

| Description |
|---|
| CAUTION: Federal law (United States) restricts this device to sale by or on<br>the order of a licensed eye care professional. |
| Steam sterlized |
| Use by date (Expiry date) |
| Batch code |
| Do not reuse |
| Do not use if bilister package is damaged |
| Example of two letter language code (English) |
| Diameter |
| Base curve |
| Power |
| Diopter (Jens power) |
| Addition power |
| European conformity sign |
| Caution |
| See product instructions |
| Authorized Representative European Community |
| Manufacturer |
| Packaging waste license sign |

a trademark of Novartis © 2016 Novartis

Manufacturer: Alcon Laboratories, Inc. 6201 South Freey Fort Worth, TX, USA 76134-2099 1-800-241-5999

March 2016

900038292-0316

- <sup>1</sup> Check for actual product availability as additional parameters may be
- introduced over time
  2 Schein, OD, Glynn RJ, Poggio EC, Seddon JM, Kenyon KR. The Relative Risk
  of Ulcerative Keratitis Among Users of Dally Wear and Extended Wear Soft
  Contact Jenses, N Eng J Med, 1989; 32321 (12):773-783



This page intentionally left blank

This page intentionally left blank



Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX 76134-2099, USA

© 2016 Novartis
\*a trademark of Novartis

March 2016

32

www.alcon.com W900087400-0316

APPENDIX I: C-QUANT STRAYLIGHT MEASUREMENT













APPENDIX J: VISIONIX CORNEAL TOPOGRAPHY AND WAVEFRONT

















# APPENDIX K:

- LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS
- EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING
- DETERMINATION OF NEAR ADDITION
- NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE
- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIVE ERROR
- BIOMICROSCOPY SCALE
- DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION
- DISTANCE LOGMAR VISUAL ACUITY MEASURMENT PROCEDURE
- PATIENT REPORTED OUTCOMES
- VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS











EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING

Title: **Expanded Sodium Fluorescein Corneal Staining Document Type: Document Number: Revision Number: 5**  Title: **Expanded Sodium Fluorescein Corneal Staining Document Type: Document Number: Revision Number: 5**
Title: Expanded Sodium Fluorescein Corneal Staining

Document Type: Revision Number: 5

#### DETERMINATION OF NEAR ADDITION

NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE

LENS FITTING CHARACTERISTICS

Title: Lens Fitting Characteristics

Document Type:
Document Number:

Revision Number: 5

SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS

DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIVE ERROR



BIOMICROSCOPY SCALE







Title: **Biomicroscopy Scale Document Type: Revision Number: 9 Document Number:** 


Title: **Biomicroscopy Scale Document Type: Revision Number: 9 Document Number:** 



#### DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION

Title: **Distance and Near Snellen Visual Acuity Evaluation Document Type: Document Number: Revision Number: 4**
DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE



| _Title: | Distance LogMAR Visual Acuity Measurement Procedure | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 4 |





## PATIENT REPORTED OUTCOMES

| Title: Document Type: Document Number: | Patient Reported Outcomes | Revision Number: | 2 |
|---|---|---|---|

## VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION

**TESTING** 

Title: **Visual Acuity Chart Luminance and Room Illumination Testing Document Type: Document Number: Revision Number: 4**  Title: Visual Acuity Chart Luminance and Room Illumination Testing **Document Type: Document Number: Revision Number: 4**  Title: Visual Acuity Chart Luminance and Room Illumination Testing

Document Type:

Document Number: 4

APPENDIX L: GUIDELINES FOR COVID-19 RISK MITIGATION

| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | · |
| <b>Document Number:</b> | | Revision Number: 4 |

#### 1.0 PURPOSE

The purpose of this document is to provide guidelines for the re-opening or initiation of clinical study sites participating in Johnson & Johnson Vision Care, Inc. (JJVCI) clinical studies during the COVID-19 pandemic.

#### 2.0 SCOPE

This document provides guidelines for Johnson & Johnson Vision Care (JJVCI) to address the potential risks from COVID-19 to study subjects, investigators, study site staff, and monitors at study sites. The guidance provided in this document is in effect from the date of approval through the date of retirement of this Work Instruction. At a minimum, this Work Instruction will be reviewed and updated on a quarterly basis, as appropriate.

NOTE: Re-opening of sites outside of the US will be evaluated on a country by country basis subject to local health authority guidance.

## 3.0 **DEFINITIONS**

American Academy of Optometry (AAO): The American Academy of Optometry is an organization of optometrists based in Orlando, Florida. Its goal is to maintain and enhance excellence in optometric practice, by both promoting research and the dissemination of knowledge. The AAO holds an annual meeting, publishes a monthly scientific journal, gives credentials to optometrists through the fellowship process and publishes position statements.

American Optometric Association (AOA): The American Optometric Association, founded in 1898, is the leading authority on quality care and an advocate for our nation's health, representing more than 44,000 Doctors of Optometry (O.D.), optometric professionals, and optometry students. Doctor of Optometry take a leading role in patient care with respect to eye and vision care, as well as general health and well-being. As primary health care providers, Doctor of Optometry have extensive, ongoing training to examine, diagnose, treat and manage ocular disorders, diseases and injuries and systemic diseases that manifest in the eye. The American Optometric Association is a federation of state, student, and armed forces optometric associations. Through these affiliations, the AOA serves members consisting of optometrists, students of optometry, paraoptometric assistants and technicians. The AOA and its affiliates work to provide the public with quality vision and eye care.

**Centers for Disease Control and Prevention (CDC):** The Centers for Disease Control and Prevention is a national public health institute in the United States. It is a United States federal agency, under the Department of Health and Human Services, and is headquartered in Atlanta, Georgia.

**COVID-19:** Current outbreak of respiratory disease caused by a novel coronavirus. The virus has been named "SARS-CoV-2" and the disease it causes has been named "Coronavirus Disease 2019" (COVID-19).

Clinical Study: Voluntary research studies conducted in people and designed to answer specific questions about the safety or effectiveness of drugs, vaccines, other therapies, or new ways of using existing treatments. May also be called clinical trials, studies, research, trials, or protocols.

Clinical Study Site: Location where a clinical study is conducted, such as a doctor's office, university, or laboratory. Clinical studies are conducted by Investigators who are individual(s) responsible for the conduct of the clinical study at a study site. If a study is conducted by a team of individuals, the Investigator is the responsible leader of the team and may be called the Principal Investigator.

**Clinical Operations Manager (COM):** The Johnson & Johnson Vision Care (JJVCI) individual responsible for the overall management of a clinical trial.


| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | |
| Document Number: | | Revision Number: 4 |

**Monitor:** An individual designated to oversee the progress of a clinical study and ensure that it is conducted, recorded, and reported in accordance with the protocol, Standard Operating Procedures (SOPs), Good Clinical Practice (GCP), and applicable regulatory requirements.

**Medical Safety Officer (MSO):** Physician who has primary accountability in their product portfolio for product health and safety, and who serves as an independent medical voice for patient safety.

**Safety Management Team (SMT):** A cross-functional, collaborative team responsible for review, assessment and evaluation of medical safety data arising from any source throughout the product life cycle.

#### 4.0 GUIDANCE FOR STUDY DOCUMENTS

In alignment with recent health authority guidance, JJVCI is providing recommendations for study-related management in the event of disruption to the conduct of the clinical study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health, safety and well-being of participants and site staff. If, at any time, a participant's safety is considered to be at risk, study intervention will be discontinued, and study follow-up will be conducted as outlined in the protocol.

During the COVID-19 pandemic, the additional risks listed below need to be considered for study participants and study personnel:

## 4.1 Additional Risks Related to the COVID-19 Pandemic:

- The possible transmission of the Coronavirus infection and consequent complications, beyond the risk of adverse events due to the investigational device and/or procedures.
- The risk may be higher in an optometric clinical study because of the close contact the subject will have with health care professionals during the procedures and assessments (since the investigator must make the measurements close to the subject's face) and, in addition the need for multiple follow-up visits/exams which may expose the subject to other patients and/or healthcare professionals who might be transmitting the virus, even if they do not have symptoms.
- Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions, which may lead to delays in scheduled follow-up visits.
- Subjects experiencing an adverse event related to contact lens wear may receive delayed treatment
  due to COVID-19 restrictions. In this event, all assessments that can be conducted virtually will be
  completed by the investigator to determine the best course of treatment for the subject, including
  an unscheduled visit, up to discontinuation from the study, as appropriate.

If a study subject is found to have contracted COVID-19 during participation in a study, he/she will be discontinued from the study and followed until COVID-19 Adverse Event (AE) resolution.

To help minimize the above potential risks, JJVCI recommend reviewing/complying with local, state, and governmental guidance for COVID-19 risks.

JJVCI will provide the following study specific documents with language pertaining to COVID-19 risks:

#### 4.1.1 Informed Consent:

Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed Consent document:


| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | |
| <b>Document Number:</b> | | Revision Number: 4 |

#### STUDY ASSOCIATED RISKS RELATED TO COVID-19 (CORONAVIRUS) PANDEMIC

It is important to note that this study will be conducted, at least in part, during the COVID-19 pandemic. As such, additional risks associated with the infection with COVID-19 exist for you. This is particularly important for this study due, in part, to the closeness of the doctor during the study examinations.

The potential effects of the disease are not fully known, at this time, and may include long-term serious health consequences. In severe cases, this may result in hospitalization and/or death. Based on current knowledge from the Centers for Disease Control and Prevention (CDC), those at high-risk for severe illness from COVID-19 include older adults and people with underlying medical conditions.

During this study, all appropriate measures will be taken to minimize risks including the use of personal protective equipment such as masks and gloves, as well as proper sanitization. This is in conformance to guidance from the CDC, local health departments, and the state and county in which the study doctor's office is located. However, these measures may not completely eliminate the risks associated with contracting COVID-19.

If you are found to have contracted COVID-19 or feel ill with flu-like symptoms during participation in the study, you will not be permitted to continue in-office study follow-up visits, but you will receive instructions and your condition will be monitored by the doctor and/or study staff.

## 4.1.2 COVID-19 Risk Control Checklist:

Will include COVID-19 risk control methods that are required by a site to conduct JJVCI clinical studies. The risk controls are consistent with CDC, AOA, AAO Guidance. The Principle Investigator will review/sign the study specific checklist prior to the Site Initiation Meeting.

Study Number Site Number Principal Investigator (PI) Name

The following COVID-19 risk control methods are required to conduct Johnson & Johnson Vison Care clinical studies. Please review the following requirements and Initial each requirement.

| PI Initials | General Site Safety Planning Measures |
|---|---|
| | Signage within site describing Risk Control methods |
| | Social Distancing practices throughout site (waiting rooms, lobby, exam rooms, etc.) |
| | Non-contact thermometer available to assess temperatures of staff and patients |
| | Training on patient flow and physical distancing in waiting room |
| | Establish longer time frame between patient appointments to reduce persons in the site |
| | Staff should receive job-specific training on PPE and demonstrate competency with selection and |
| | proper use of PPE and wear at all times during interactions with subjects (e.g., putting on and |
| | removing without self-contamination) |

| PI Initials | Site Staff Daily Safety Measures |
|---|---|
| | As part of routine practice, site staff should regularly monitor themselves for fever and symptoms |
| | of COVID-19, including temperature checks |
| | Any staff member (including Investigators) showing signs of being sick or testing positive for |
| | COVID-19 should not be permitted to work and the Sponsor shall be informed |
| | NOTE: Inform JJVC in 24 hours of any significant impact to the study. |
| | Ensure that all staff wear a mask |
| | Gloves should be required when working directly with patients and changed between each patient |


| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | |
| <b>Document Number:</b> | Revision Numb | er: 4 |
| | Have staff thoroughly wash hands for at least 20 seconds or use an alcohol-based hand sanitizer | |
| | when they arrive, before and after each patient, before eating and after using the bathroom. | |
| | Cleaning and disinfection procedures for exam rooms and instruments or equipment between | |

Cleaning and disinfection procedures for commonly touched surfaces (doors, chairs, computers,

| PI Initials | Before a Patient or Study Visit: |
|---|---|
| | Patients should be asked prior to entering the site about fever and respiratory illness and whether |
| | they or a family member have had contact with another person with confirmed COVID-19 in the |
| | past 14 days. Patients exhibiting signs of being sick should be rescheduled when their symptoms |
| | resolve. |
| | Instruct patients that companions should remain outside of the facility and not accompany the patient into the facility unless they are a parent/guardian of the patient or if they are a true |
| | caregiver and need to assist the patient |
| | Request the patient to call or text the office upon arrival so entrance to and movement through |
| | facility can be coordinated by site staff |

| PI Initials | Patients Entering the site: |
|---|---|
| | Temperature checks utilizing a non-contact thermometer for all patients and companions entering |
| | the site. |
| | All patients and companions must wear cloth or disposable mask at all times in the site |
| | Maintain social distancing. Waiting rooms or lobbies should be as empty as possible. Advise |
| | seated patients to remain at least 6 feet from one another. |
| | Communal objects in (e.g. toys, reading materials, etc.) should be removed or cleaned regularly. |

I certify that I have read and agree to implement all the listed COVID-19 Risk Control Measures required for the conduct of Johnson & Johnson Vision Care studies.

Principal Investigator Signature and Date

patients with gloves.

phones, etc.) with gloves.


| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | |
| Document Number: | | Revision Number: 4 |

## RESOURCE LINKS

## **US Resource Links**

OSHA Training

https://www.osha.gov/SLTC/covid-19/controlprevention.html

Personal Protective Equipment (PPE) Training

CDC: https://www.cdc.gov/coronavirus/2019-ncov/hcp/using-ppe.html

I&R Training

ACUVUE® LensAssist: https://www.acuvue.com/lensassist

• Clinic Preparedness Guides

CDC: <a href="https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinic-preparedness.html">https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinic-preparedness.html</a>
AOA: <a href="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://www.aoa.org/optometry-practice-reactivation-preparedness-guide">https://www.aoa.org/optometry-practice-reactivation-preparedness-guide</a>

• In-Office Disinfection of Multi-Patient Use Diagnostic Contact Lenses

<a href="https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnostic-lenses.pdf">https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnostic-lenses.pdf</a>

## **OUS Resource Links**

- Updates on local regulations in Hong Kong https://www.coronavirus.gov.hk/eng/index.html
- Resumption of optical services in England: Letter from Matt Neligan and Poonam Sharma
   <a href="https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-optical-services-letter-17-june-2020.pdf">https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-optical-services-letter-17-june-2020.pdf</a>
- NHS Optical Letter
   <a href="https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf">https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf</a>
- The College of Optometrists primary eye care COVID-19 guidance: Red phase
   <a href="https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html">https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html</a>
  <a href="https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html">https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html</a>
- The College of Optometrists COVID-19: College updates https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-2019-advice-for-optometrists.html#CollegeGuidelines
- Infection Control Guidelines. (n.d.). Retrieved from Canadian Association Of Optometrists: https://opto.ca/sites/default/files/resources/documents/infection\_control\_guidelines\_2016.pdf
- Infection prevention and control for COVID-19: Interim guidance for outpatient and ambulatory care settings. (2020, May 23 May). Retrieved from Government of Canada: https://www.canada.ca/en/public-health/services/diseases/2019-novel-coronavirus-infection/guidance-documents/interim-guidance-outpatient-ambulatory-care-settings.html


| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | |
| <b>Document Number:</b> | | <b>Revision Number: 4</b> |

• Information for Members On Coronavirus (COVID-19). (n.d.). Retrieved from Canadian Association Of Optometrists:

 $https://opto.ca/sites/default/files/resources/documents/information\_for\_members\_on\_coronavirus.pdf$ 

 Coronavirus (COVID-19) resources for health professionals, including aged care providers, pathology providers and health care managers. (2020, September 24). Retrieved from Australian Government Department of Health:

https://www.health.gov.au/resources/collections/coronavirus-covid-19-resources-for-health-professionals-including-aged-care-providers-pathology-providers-and-health-care-managers

- Environmental Cleaning and Disinfection Principles for COVID-19. (n.d.). Retrieved from Australian Government Department of Health:
  - https://www.health.gov.au/sites/default/files/documents/2020/03/environmental-cleaning-and-disinfection-principles-for-covid-19.pdf
- Infection control guidelines and advice. (n.d.). Retrieved from Optometry Australia: https://www.optometry.org.au/practice-professional-support/coronavirus-covid-19-what-optometrists-need-to-know/covid-19-clinical-advice/infection-control-guidelines-and-advice/

## 4.1.3 Protocol Compliance Investigator(s) Signature Page:

Will include a statement indicating that the Principal Investigator (PI) agrees to conduct the study in compliance with all local, state, and governmental guidance's for COVID-19 risk mitigation.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

4.1.4 Study Site Initiation Training Slides:

Will include suggestions to help mitigate potential transmission of COVID-19. Suggestions may include maintaining social distancing in the clinical site by staggered scheduling of study patients, wearing proper PPEs, frequent disinfection, and installing shields on the slit lamp and other applicable equipment.

## 5.0 GUIDANCE FOR REMOTE SUBJECT VISITS

Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions. Possible disruption of the study as a result of COVID-19 control measures may lead to delays in scheduled follow-up visits.

Subjects may be delayed in being seen for study follow up visit(s), for example due to COVID-19 control measures or due to the subject's concerns or fears about COVID-19 risk. When appropriate, the remote assessment will be conducted to the extent possible. Discussions with the subject during remote assessments may include:


| Title: | <b>Guidelines for COVID-19 Risk Mitigation</b> |
|--------|------------------------------------------------|
|--------|------------------------------------------------|

| Document Type: | Work Instruction | |
|-----------------|------------------|--------------------|
| Document Number | VWI_0081 | Revision Number: 4 |

| Procedure | Details |
|---|---|
| Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire regarding the test article when applicable and feasible. |
| Change of Medical History<br>(Adverse Events) and<br>Concomitant Medications /<br>Therapies Review | Record any adverse events or medical history changes from the previous study visit with the subject/parents. Review the subject's concomitant medications/therapies and record any changes from the previous study visit. |
| Wearing Time and Compliance | Record the average wearing time (including number of hours per day during weekdays and weekends, and number of days per week). Confirm compliance with the prescribed wear schedule. Record and discuss the lens wear compliance based on the subject's self-report. For example, the subjects will be asked the time of the day the subject typically puts on the study lenses in the morning and takes off in the evening, the number of days per week lenses were worn, and the number of consecutive days the subject didn't wear the study lenses, etc. |

The discussion with the subject will be documented in EDC under Tele-Visit and a minor protocol deviation will be noted. If during the telephone consultation, a subject states he/she wishes to discontinue participating in the study, instruct the subject to stop wearing the study lenses and schedule the subject to return to the clinic for a Final Evaluation at the at earliest possible time. Subjects should return all unused lenses to the clinic at the last visit.

Changes in study visit schedules, missed visits, or participant discontinuations may lead to missing data, including data related to protocol-specified procedures. Case report forms should capture specific information regarding the basis of missing data, including the relationship to the COVID-19 pandemic.

#### 6.0 STUDY CONDUCT DURING PANDEMIC

It is recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantine by participants and study-site personnel; travel restrictions/limited access to public places, including Optometry Clinics; and changes in clinic procedures required to address the COVID-19 challenge.

Every effort should be made to adhere to protocol-specified assessments for study participants, including follow-up. However, if scheduled visits cannot be conducted in person at the study site it is suggested that assessments be performed to the extent possible remotely/virtually or delayed until such time that on-site visits can be resumed in order to continue participant monitoring in accordance with the protocol where possible. At each contact, participants will be interviewed to collect safety data. Key efficacy endpoint assessments should be performed if required and as feasible.

Modifications to protocol-required assessments may be permitted via COVID-19 Appendix after consultation with the participant, investigator, and the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol deviations. Interruptions of test article wear or discontinuations of study interventions and withdrawal from the study should be documented with the prefix "COVID-19-related" in the case report form (CRF).


| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | · |
| Document Number: | | Revision Number: 4 |

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to local guidance.

If a participant has tested positive for COVID-19, the investigator should contact the sponsor's responsible medical monitor to discuss initial plans for study intervention and follow-up. The medical monitor will notify the Safety Management Team of any subject(s) that have reported "COVID-19", "Asymptomatic COVID-19", or "Suspected COVID-19" adverse events within 24 hours of the notification.

Modifications made to the study conduct as a result of the COVID-19 pandemic will be summarized in the clinical study report.

COVID-19 screening procedures that may be mandated by local healthcare systems do not need to be reported as an amendment to the protocol even if done during clinical study visits.

## 6.1 Monitoring Visits

When on-site monitoring by the sponsor is not feasible, the sponsor's site monitor will contact the study site to schedule remote visits. In such cases, on-site monitoring visits will resume when feasible, with increased frequency to address the source data verification backlog.

Even with staffing limitations during this COVID-19 pandemic, all routine operations related to clinical trials should be well-documented and archived as part of standard process. When conditions permit, all parties involved in this clinical trial should communicate relevant information in a timely manner so that all relevant parties remain sufficiently informed.

#### 6.1.1 Study Site Initiation:

During the period that this Work Instruction is in effect, Site Initiation Meetings and training of study site staff will be conducted remotely. The JJVCI study team will conduct training via Skype, Zoom, Microsoft Teams or similar software as well as utilize online training materials, as applicable. Study site training will be documented utilizing Site Initiation Report

On-site visits may be considered when, for example, hands-on training or evaluation of site facilities is required. While on site, the Clinical Research Associate (CRA) will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

## 6.1.2 Interim Monitoring Visits (if applicable):

During the period that this Work Instruction is in effect, Interim Monitoring On-site visits will be kept to a minimum and include only those tasks that the CRA cannot perform remotely (e.g., source document verification, test article reconciliation, etc.).

To ensure data integrity during the conduct of all JJVC studies, clinical study teams will follow the study specific Clinical Monitoring Plan

While on site, the CRA will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.


| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | |
| <b>Document Number:</b> | | Revision Number: 4 |

## 6.1.3 Study Site Closure:

During the period that this Work Instruction is in effect, the duration of the Study Site Closure Visit will be limited to tasks that the CRA cannot perform remotely (e.g., source document verification, test article final reconciliation and return, etc.).


| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | Work Instruction | |
| <b>Document Number:</b> | | Revision Number: 4 |

## **Attachment A: Study Site Correspondence**

XXXX XX, 2020

## Re: COVID-19 Mitigation Plan, <<CR-xxxx/protocol title>>

Dear << Principal Investigator>> and Study Team,

Coronavirus (COVID-19) has impacted several communities and business activities over the past several months. While we work toward the successful conduct of clinical studies, our commitment continues to be the safety of patients, healthcare professionals, and to our communities.

Therefore, we would like to share the following revisions/additions related to the above referenced Johnson & Johnson Vision Care company sponsored clinical trial(s) you are currently working on or considering participation within.

## **Protocol:**

• Guidelines for COVID-19 Risk Mitigation provided in the Appendix section.

## **Protocol Signature Page:**

 Will include a statement indicating the Principle Investigator agrees to conduct the study in compliance with all local, state, and governmental guidelines for COVID-19 risk mitigation.

## **Informed Consent:**

• Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed consent document.

## **COVID-19 Risk Control Checklist for Clinical Studies:**

• Will include COVID-19 risk control measures that are required to ensure the safety and health of subjects, site staff and monitors during the pandemic.

We want to encourage the need for open lines of communication about potential challenges you may foresee as the result of the current COVID-19 situation. Therefore, we encourage you to regularly connect with your respective Johnson & Johnson clinical study team (Clinical Research Associate (CRA), Lead CRA or Study Managers).

Thank you for your continued engagement, collaboration, and dedication to your study subjects during this challenging time.

Please file this letter in your site file study correspondence.


## PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6418 Evaluation of Investigational Daily Disposable Multifocal Contact Lenses Produced with Different Manufacturing Processes

Version and Date: 2.0 10 February 2021

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

| Principal<br>Investigator: | | |
|----------------------------|------------------------------------------|------|
| _ | Signature | Date |
| Institution/Site: | Name and Professional Position (Printed) | _ |
| | Institution/Site Name | |
| | Institution/Site Address | |